

### STATISTICAL ANALYSIS PLAN

Study Title: A Phase 3, Randomized, Open Label Study to Evaluate the Safety

and Efficacy of Switching to a Fixed Dose Combination (FDC) of GS-9883/Emtricitabine/Tenofovir Alafenamide (GS-9883/F/TAF)

from Elvitegravir/Cobicistat/Emtricitabine/

Tenofovir Alafenamide (E/C/F/TAF), Elvitegravir/Cobicistat/ Emtricitabine/Tenofovir Disoproxil Fumarate (E/C/F/TDF) or Atazanavir + Ritonavir + Emtricitabine/Tenofovir Disoproxil Fumarate (ATV+RTV+FTC/TDF) in Virologically Suppressed

HIV-1 Infected Women

Name of Test Drug: Bictegravir/Emtricitabine/Tenofovir Alafenamide (B/F/TAF;

GS-9883/F/TAF)

Study Number: GS-US-380-1961

Protocol Version (Date): Amendment 2 (10 November 2016)

Analysis Type: Week 48 Interim Analysis

Analysis Plan Version: Version 1.0

Analysis Plan Date: 19 October 2017

Analysis Plan Author(s): PPD

CONFIDENTIAL AND PROPRIETARY INFORMATION

## **TABLE OF CONTENTS**

| TAI | BLE OF | F CONTENTS | 2 |
|---|---|---|---|
| LIS | T OF T | ABLES | 4 |
| LIS | T OF A | BBREVIATIONS | 5 |
| 1. | INTR | ODUCTION | 8 |
| | 1.1. | Study Objectives | |
| | 1.1. | Study Design | |
| | 1.3. | Sample Size and Power | |
| 2. | TYPE | OF PLANNED ANALYSIS | |
| | 2.1. | Data Monitoring Committee Analysis | 11 |
| | 2.2. | Week 48 Interim Analysis | |
| | 2.3. | Final Analysis | 11 |
| 3. | GENE | ERAL CONSIDERATIONS FOR DATA ANALYSES | 12 |
| | 3.1. | Analysis Sets | 13 |
| | | 3.1.1. All Randomized Analysis Set | 13 |
| | | 3.1.2. Full Analysis Set | |
| | | 3.1.3. Per Protocol Analysis Set | |
| | | 3.1.4. Safety Analysis Set | |
| | | 3.1.5. Pharmacokinetic (PK) Analysis Set | |
| | 3.2. | Subject Grouping | |
| | 3.3. | Strata and Covariates. | |
| | 3.4. | Examination of Subject Subgroups | |
| | | 3.4.1. Subject Subgroups for Efficacy Analyses | |
| | 3.5. | 3.4.2. Subject Subgroups for Safety Analyses | |
| | 3.6. | Missing Data and Outliers | |
| | 3.0. | 3.6.1. Missing Data | |
| | | 3.6.2. Outliers | |
| | 3.7. | Data Handling Conventions and Transformations | |
| | 3.8. | Analysis Windows | |
| | | 3.8.1. Definition of Study Day | 18 |
| | | 3.8.2. Analysis Windows | 19 |
| | | 3.8.3. Selection of Data in the Event of Multiple Records in an Analysis | |
| | | Window | 21 |
| 4. | SUBJ | ECT DISPOSITION | |
| | 4.1. | Subject Enrollment and Disposition | 22 |
| | | 4.1.1. Subject Enrollment | |
| | 4.0 | 4.1.2. Subject Disposition | |
| | 4.2. | Extent of Study Drug Exposure and Adherence. | |
| | | 4.2.1. Duration of Exposure to Randomized Study Drug | |
| | 4.3. | 4.2.2. Adherence to Study Drug Regimen | |
| 5. | BASE | LINE CHARACTERISTICS | 26 |
| | 5.1. | Demographics and Baseline Characteristics | 26 |
| | 5.2. | Baseline Disease Characteristics | |
| | 5.3 | Medical History | 27 |

| 6. | EFFI | ICACY ANALYSES | 28 |
|---|---|---|---|
| | 6.1. | Primary Efficacy Endpoint | 28 |
| | | 6.1.1. Definition of the Primary Efficacy Endpoint | 28 |
| | | 6.1.2. US FDA-defined Snapshot Algorithm | |
| | | 6.1.3. Statistical Hypothesis for the Primary Efficacy Endpoint | 29 |
| | | 6.1.4. Primary Analysis of the Primary Efficacy Endpoint | 29 |
| | | 6.1.5. Secondary Analysis of the Primary Efficacy Endpoint | |
| | 6.2. | Secondary Efficacy Endpoints | 30 |
| | | 6.2.1. Definition of the Secondary Efficacy Endpoints | |
| | | 6.2.2. Analysis of the Secondary Efficacy Endpoints | |
| | 6.3. | Tertiary Efficacy Endpoints | |
| | | 6.3.1. Definition of the Tertiary Efficacy Endpoints | |
| | <i>C</i> 1 | 6.3.2. Analysis of the Tertiary Efficacy Endpoints | |
| | 6.4. | Changes From Protocol-Specified Efficacy Analyses | |
| 7. | SAFE | ETY ANALYSES | |
| | 7.1. | Adverse Events and Deaths | |
| | | 7.1.1. Adverse Event Dictionary | |
| | | 7.1.2. Adverse Event Severity | |
| | | 7.1.3. Relationship of Adverse Events to Study Drug | |
| | | 7.1.4. Serious Adverse Events | |
| | | 7.1.5. Treatment-Emergent Adverse Events | |
| | | 7.1.6. Summaries of Adverse Events and Death | |
| | 7.2. | 7.1.7. Additional Analysis of Adverse Events | |
| | 1.2. | 7.2.1. Summaries of Numeric Laboratory Results | |
| | | 7.2.1. Summaries of Numeric Laboratory Results | |
| | | 7.2.3. Metabolic Laboratory Evaluations | |
| | | 7.2.4. Liver-Related Laboratory Evaluations | |
| | | 7.2.5. Renal-Related Laboratory Evaluations | |
| | 7.3. | Body Weight, Height, and Vital Signs | |
| | 7.4. | Prior and Concomitant Medications | |
| | | 7.4.1. Antiretroviral Medications | |
| | | 7.4.2. Prior Antiretroviral Medications | |
| | | 7.4.3. Concomitant Non-Antiretroviral Medications | 44 |
| | 7.5. | Electrocardiogram Results | |
| | 7.6. | Other Safety Measures | |
| | 7.7. | Subject Subgroup for Safety Endpoints | |
| | 7.8. | Changes From Protocol-Specified Safety Analyses | 45 |
| 8. | PHAI | RMACOKINETIC ANALYSES | 46 |
| | 8.1. | Analysis for Trough and Postdose PK (PK Analysis Set) | 46 |
| | 8.2. | Changes from Protocol-Specified Pharmacokinetic Analysis | |
| 9. | SPEC | CIAL POPULATION ANALYSES | 47 |
| | 9.1. | Analyses for HIV/HBV Coinfected Subjects | 47 |
| | 9.2. | Analyses for HIV/HCV Coinfected Subjects | |
| 10. | REFE | ERENCES | 50 |
| 11. | SOFT | TWARE | 51 |
| 12. | SAP REVISION5 | | |
| 13. | APPENDICES 5 | | |

| Appendix 1. Appendix 2. Appendix 3. Appendix 4. Appendix 5. | Study Procedures Table Flowchart of US FDA-defined Snapshot Algorithm Selected Medical History Hepatic Events Programming Specification | 58<br>7 |
|---|---|---|
| | LIST OF TABLES | |
| Table 3-1. | Subjects Excluded from Week 48 PP Analysis Set Due to Premature Discontinuation of Study Drug and/or Missing HIV-1 RNA Assessment in Week 48 Analysis Window | 14 |
| Table 3-2. | Analysis Windows for HIV-1 RNA, CD4+ cell count, CD4 %, HBV DNA, Hematology, Chemistry, Urinalysis, and Urine Pregnancy Laboratory Tests, eGFR <sub>CG</sub> , Vital Signs, and Weight | |
| Table 3-3. | Analysis Windows for Metabolic Assessments and HBV Serology | |
| Table 3-4. | Analysis Windows for TSH, Renal Function, and Safety ECG | |
| Table 3-5. | Analysis Windows for HCV Serology and HCV RNA Assessments | |

### LIST OF ABBREVIATIONS

AE adverse event

ALP alkaline phosphatase
ALT alanine aminotransferase
ANOVA analysis of variance

ARV antiretroviral

AST aspartate aminotransferase

ATV Atazanavir

B2M beta-2 microglobulin
BIC Bictegravir, GS-9883, B

B/F/TAF single-tablet regimen of bictegravir (BIC; B) 50 mg / emtricitabine (FTC) 200 mg /

tenofovir alafenamide (TAF) 10 mg; GS-9883/F/TAF

BLQ below limit of quantitation

BMI body mass index
BSA body surface area
CG Cockroft-Gault
CI confidence interval

CMH Cochran-Mantel-Haenszel

CRF case report form
CSR clinical study report
DNA Deoxyribonucleic Acid

DOB date of birth

DSPH Drug Safety and Public Health Department

E/C/F/TAF Elvitegravir /Cobicistat /Emtricitabine/ Tenofovir Alafenamide; Genvoya; GEN E/C/F/TDF Elvitegravir /Cobicistat /Emtricitabine / Tenofovir Disoproxil Fumarate; Stribild;

STB

ECG electrocardiogram

eCRF electronic case report form

eGFR estimated glomerular filtration rate

eGFR(CG) estimated glomerular filtration rate using Cockcroft-Gault formula

FAS full analysis set

FDA Food and Drug Administration

FDC fixed dose combination

FTC/TDF single-tablet regimen of emtricitabine 200 mg/ tenofovir alafenamide 10 mg

FTC Emtricitabine: F

GFR glomerular filtration rate
GGT gamma-glutamyl transferase

Gilead Gilead Sciences, Inc.
GS-9883 Bictegravir; BIC; B
HBcAb hepatitis B core antibody

HBeAb hepatitis B e-antibody
HBeAg hepatitis B e-antigen

HBsAb hepatitis B surface antibody HBsAg hepatitis B surface antigen

HBV hepatitis B virus
HCV hepatitis C virus
HCVAb HCV antibody

HDL high density lipoprotein

HIV-1 human immunodeficiency virus (Type 1)

HLGT high level group term
HLT high level term
ID identification

IDMC independent data monitoring committee

INR international normalized ratio
IWRS interactive web response system

KM Kaplan-Meier

LDL low density lipoprotein LLOQ lower limit of quantitation

LLT lowest level term

LOCF last observation carried forward

MedDRA Medical Dictionary for Regulatory Activities

MH Mantel-Haenszel
OLE open-label extension
PK pharmacokinetic
PP per protocol
PT preferred term
PT prothrombin time

Q quartile
Q1 first quartile
Q3 third quartile

RBP retinol binding protein
RNA ribonucleic acid

RTV Ritonavir

SAE serious adverse events
SAP statistical analysis plan
SBR stay on baseline regimen

SD standard deviation SE standard error

SMQ Standardised MedDRA Query

SOC system organ class

TAF tenofovir alafenamide
TEAE treatment-emergent AE
TFL tables, figures, and listings

TFV tenofovir

TSH thyroid stimulating hormone

ULN upper limit of normal

UACR urine albumin to creatinine ratio
WHO World Health Organization

### 1. INTRODUCTION

This statistical analysis plan (SAP) describes the statistical analysis methods and data presentations to be used in tables, figures, and listings (TFLs) of the Week 48 interim analysis for Study GS-US-380-1961, which will be performed when all subjects have completed their Week 48 visit or prematurely discontinued from the study drug. This SAP is based on the study protocol amendment 2 dated 10 November 2016 and the electronic case report form (eCRF). The SAP will be finalized before data finalization for the interim analysis. Any changes made after the finalization of the SAP will be documented in the clinical study report (CSR).

### 1.1. Study Objectives

The primary objective of this study is:

• To evaluate the efficacy of switching to a fixed dose combination (FDC) of bictegravir (GS-9883; BIC; B) /emtricitabine (FTC; F) /tenofovir alafenamide (TAF) versus continuing on a regimen consisting of E/C/F/TAF, E/C/F/TDF, or ATV+RTV+FTC/TDF in virologically suppressed HIV-1 infected women as determined by the proportion of subject with HIV-1 RNA ≥ 50 copies/mL at Week 48.

The secondary objective of this study is:

• To evaluate the safety and tolerability of the treatment groups through Weeks 48.

## 1.2. Study Design

#### **Design Configuration and Subject Population**

GS-US-380-1961 is a randomized, open label, multicenter, active-controlled study to evaluate the safety and efficacy of switching to an FDC of B/F/TAF in HIV-1 infected women who are virologically suppressed (HIV-1 RNA < 50 copies/mL) on a regimen consisting of E/C/F/TAF, E/C/F/TDF, or ATV+RTV+FTC/TDF for  $\geq$  12 consecutive weeks prior to screening.

All subjects will be HIV-1 infected women drawn from pre-defined Gilead Sciences In. (Gilead) clinical studies and must be virologically suppressed. Women in Gilead study GS-US-236-0128 who completed the Week 48 open-label extension (OLE) visit or any post Week 48 OLE visits, women in study GS-US-292-0109 who completed the Week 96 visit or any post Week 96 visits, or women in studies GS-US-292-0104 or GS-US-292-0111 who completed the Week 144 visit or any post Week 144 visits may be eligible to enroll.

#### **Treatment Groups**

Subjects who provide written consent and meet all eligibility criteria will be randomized in a 1:1 ratio to receive open label medication as follows:

**Treatment Group 1:** FDC of BIC 50 mg/FTC 200 mg/TAF 25 mg (B/F/TAF) administered orally, once daily, without regard to food (approximately n = 235)

**Treatment Group 2:** Stay on baseline regimen (SBR), including E/C/F/TAF, E/C/F/TDF, or ATV+RTV+FTC/TDF administered orally, once daily, with food (approximately n = 235)

### **Key Eligibility Criteria**

Medically stable HIV-1 infected women who meet the following criteria:

- Currently on a stable antiretroviral regimen consisting of E/C/F/TAF, E/C/F/TDF, or ATV+RTV+FTC/TDF continuously for ≥ 12 consecutive weeks preceding the screening visit
- Documented plasma HIV-1 RNA levels < 50 copies/mL for ≥ 12 weeks preceding the Screening visit. After reaching HIV-1 RNA < 50 copies/mL, single values of HIV-1 RNA ≥ 50 copies/mL followed by re-suppression to < 50 copies/mL is allowed
- HIV-1 RNA <50 copies/mL at screening
- Estimated glomerular filtration rate (eGFR) ≥ 50 mL/min according to the Cockcroft-Gault (C-G) formula at the screening visit

### **Study Periods / Phases**

Subjects will be treated for at least 48 weeks. At the Week 48 Visit, subjects in a country where B/F/TAF FDC is not available will be given the option to receive B/F/TAF FDC for an additional 48 weeks, or until the product becomes accessible to subjects through an access program, or until Gilead elects to discontinue the study in that country, whichever occurs first.

Subjects who complete the study through the Week 48 Visit and do not continue participation in the study will be required to return to the clinic 30 days after the Week 48 Visit for a 30 Day Follow-Up Visit.

#### **Schedule of Assessments**

After screening procedures, eligible subjects will be randomized 1:1 to Treatment Group 1 or Treatment Group 2 and treated for 48 weeks. Following the Screening and Day 1 visits, subjects will return for study visits at Weeks 4, 8, 12, and then every 12 weeks until the Week 48 visit.

For all eligible subjects, blood and urine will be collected at Day 1, Weeks 4, 8, 12, and then every 12 weeks through the Week 48 visit. Laboratory analyses (including hematology, chemistry, and urinalysis), HIV-1 RNA, CD4+ cell count, and complete or symptom directed physical examinations will be performed at the Screening, Day 1, and all subsequent study visits.

Adverse events and concomitant medications will be assessed at each visit.

#### **Pharmacokinetics**

For all subjects on B/F/TAF (Treatment Group 1), a single anytime pre or post-dose PK blood sample will be collected at Weeks 8, 24, and 36.

For all subjects on B/F/TAF (Treatment Group 1), a trough PK blood sample will be obtained 20-28 hours following the last dose at Weeks 4 and 12. Following an observed dose, one PK blood sample will be collected between 1 and 4 hours post-dose.

The concentration of BIC may be summarized using descriptive statistics.

#### Randomization

Subjects will be randomized in a 1:1 ratio to 1 of 2 Treatment Groups (Treatment Group 1: Treatment Group 2). Randomization will be stratified by the prior treatment regimen group (ie, E/C/F/TAF, E/C/F/TDF, and ATV+RTV+FTC/TDF).

### Site and/or Stratum Enrollment Limits

Approximately 57 study sites in North America, Dominican Republic, Thailand, Russia, and Uganda participated. There was no enrollment limit for individual sites.

## **Study Duration**

The randomized phase of this study is 48 weeks in duration.

# 1.3. Sample Size and Power

A total of approximately 470 HIV-1 infected women, randomized in a 1:1 ratio to 2 treatment groups (approximately 235 subjects per treatment group), achieves at least 87% power to detect a non-inferiority margin of 4% difference in the percentage of subjects with HIV-1 RNA ≥ 50 copies/mL at Week 48 between the 2 treatment groups.

For sample size and power computation, it is assumed that both treatment groups have 2% of subjects with HIV-1 RNA  $\geq 50$  copies/mL at Week 48 (based on the historical Gilead Genvoya<sup>®</sup>[GEN; E/C/F/TAF] and Stribild<sup>®</sup> [STB; E/C/F/TDF] studies), that a non-inferiority margin is 4%, and that the significance level of the test is at a one-sided 0.025 level. Sample size and power calculations were made using the statistical software package nQuery Advisor (Version 6.0).

## 2. TYPE OF PLANNED ANALYSIS

## 2.1. Data Monitoring Committee Analysis

The Week 24 Independent Data Monitoring Committee (IDMC) analysis was conducted after all subjects enrolled completed their Week 24 visit of the study or prematurely discontinued the study drug. The purpose of this interim analysis was to provide the IDMC with a statistical report for review. More details are documented in the IDMC charter.

Gilead does not have a prior intent to ask the IDMC to review Week 48 result or to consider early termination of the study even if there is early evidence of favorable efficacy for B/F/TAF.

### 2.2. Week 48 Interim Analysis

The Week 48 interim analysis will be conducted after all subjects either complete their Week 48 visit or prematurely discontinue from the study drug.

This statistical analysis plan describes the analysis plan for the Week 48 interim analysis, the primary analysis of this study.

### 2.3. Final Analysis

The final statistical analysis will be conducted after all subjects either complete the study or prematurely discontinue from the study.

### 3. GENERAL CONSIDERATIONS FOR DATA ANALYSES

The Week 48 interim analysis will include all data collected from the randomized and the extension phases of the study. Only data collected in the randomized phase (ie, randomized phase data) will be summarized by treatment group, if not specified otherwise. Data collected from both phases will be included in data listings. Data included in each phase are defined as follows:

#### **Randomized Phase Data**

- For subjects who are never treated in the extension phase of the study, all available data are considered as the randomized phase data.
- For subjects treated in the extension phase of the study, randomized phase data are defined as data collected **up to** the extension phase first dose date except for data on adverse events (AEs), concomitant medications, pregnancy, and death. For AEs, concomitant medications, pregnancy, and death, only data collected **prior to** the extension phase first dose date are included

#### **Extension Phase Data**

 Extension phase data are only available from subjects who enter the extension phase of the study. Extension phase data are defined as data collected after the extension phase first dose date except for data on AEs, concomitant medications, pregnancy, and death. For AEs, concomitant medications, pregnancy, and death, data collected on or after the extension phase first dose date are included.

Analysis results will be presented using descriptive statistics. For categorical variables, the number and percentage of subjects in each category will be presented; for continuous variables, the number of subjects (n), mean, standard deviation (SD) or standard error (SE), median, first quartile (Q1), third quartile (Q3), minimum, and maximum will be presented.

All statistical tests will be 2-sided and performed at the 5% significance level unless otherwise specified.

By-subject listings will be presented for all subjects in the All Randomized analysis set unless otherwise specified, and sorted by subject ID number, visit date, and time (if applicable). Data collected on log forms, such as AEs, will be presented in chronological order within a subject. The treatment group to which subjects were randomized will be used in the listings.

In general, age (in years) on the date of the first dose of study drug will be used for analyses and presentation in listings. For randomized but never dosed subjects, age on the date of randomization will be used. For screen failures, age on the date of the informed consent was signed will be used. If only birth year is collected on the eCRF, "01 January" will be used for the unknown birth day and month for the purpose of age calculation, similarly, if only birth year and month are collected on the eCRF, "01" will be used for the unknown birth day for the purpose of age calculation.

In general, permanent discontinuation of the randomized study drug refers to premature discontinuation of the randomized study drug or completion of the randomized study drug. Similarly, permanent discontinuation of the extension study drug refers to premature discontinuation of the extension study drug or completion of the extension study drug.

### 3.1. Analysis Sets

Analysis sets define the subjects to be included in an analysis. Analysis sets and their definitions are provided in this section. Subjects included in each analysis set will be determined before data finalization. The analysis set will be included as a subtitle of each table, figure, and listing. A summary of the number and percentage of subjects in each analysis set will be provided by treatment group and in total.

### 3.1.1. All Randomized Analysis Set

The **All Randomized Analysis Set** will include all subjects who are randomized into the study. This is the primary analysis set for by-subject listings.

## 3.1.2. Full Analysis Set

The **Full Analysis Set (FAS)** will include all subjects who (1) are randomized into the study and (2) have received at least 1 dose of randomized study drug. Subjects will be grouped according to the treatment to which they were randomized. For the FAS, all randomized phase efficacy data will be included, unless specified otherwise. This is the primary analysis set for efficacy analyses.

### 3.1.3. Per Protocol Analysis Set

The Week 48 **Per Protocol (PP) Analysis Set** will include all subjects who (1) are randomized into the study, (2) have received at least 1 dose of randomized study drug, and (3) have not committed any major protocol violation, including the violation of key entry criteria. Subjects will be grouped according to the treatment they actually received. For the PP analysis, randomized phase efficacy data collected up to 1 day after the randomized phase last dose date will be included. The Week 48 PP analysis set is the secondary analysis set for efficacy analysis.

Subjects meeting any of the following criteria will be excluded from the Week 48 PP analysis set:

• Subjects who do not have an on-treatment HIV-1 RNA in the Week 48 analysis window, except when missing is due to discontinuation of study drug for lack of efficacy. (Note: lack of efficacy is defined as having the check-box for Lack of Efficacy marked as the reason for premature study drug discontinuation on the Randomized Phase Study Drug Completion eCRF page; Table 3-1).

Table 3-1. Subjects Excluded from Week 48 PP Analysis Set Due to Premature Discontinuation of Study Drug and/or Missing HIV-1 RNA Assessment in Week 48 Analysis Window

| Discontinuation from Study Drug prior to or on the<br>Upper Bound of Week 48 Analysis Window | | HIV-1 RNA Data on Randomized Treatment<br>Available in Week 48 Analysis Window | |
|---|---|---|---|
| | | Yes | No |
| Vac | Due to Lack of Efficacy | + | + |
| Yes | Due to Other Reasons | + | - |
| No | | + | - |

<sup>+ =</sup> Inclusion of Subjects in Week 48 PP analysis set; - = Exclusion of Subjects in Week 48 PP analysis set.

- Subjects who do not meet the inclusion criteria for no documented or suspected resistance to FTC, TFV, ATV, or EVG, including but not limited to the reverse transcriptase resistance mutations K65R and M184V/I.
- Subjects who meet the exclusion criterion for receiving ongoing therapy with any of the medications listed in Tables 5-1 and 5-2 in protocol Section 5.4.
- Nonadherence to study drug: subjects with adherence rate for active study drug up to the Week 48 Visit below the 2.5th percentile.

## 3.1.4. Safety Analysis Set

The **Safety Analysis Set** will include all subjects who (1) are randomized into the study and (2) have received at least 1 dose of randomized study drug. All randomized phase safety data collected up to 30 days from the randomized phase last dose date will be included in the safety summaries, unless specified otherwise. Subjects will be grouped according to the treatment they actually received. This is the primary analysis set for safety analyses.

#### 3.1.5. Pharmacokinetic (PK) Analysis Set

The **PK Analysis Set** will include all subjects who (1) are randomized into the B/F/TAF treatment group, (2) have received at least 1 dose of B/F/TAF in the randomized phase of the study, and (3) have at least 1 nonmissing PK concentration value for any analyte of interest reported by the PK lab. The PK analysis set will be used for general PK analyses.

## 3.2. Subject Grouping

For analyses based on the All Randomized Analysis Set or the FAS, subjects will be grouped by randomized treatment. For other analyses, subjects will be grouped by actual treatment received. The actual treatment received will differ from the randomized treatment only when the actual treatment received differs from randomized treatment for the entire treatment duration.

### 3.3. Strata and Covariates

There is no stratification for analysis.

## 3.4. Examination of Subject Subgroups

## 3.4.1. Subject Subgroups for Efficacy Analyses

The proportion of subjects with HIV-1 RNA < 50 copies/mL at Week 48 as determined by the US FDA-defined snapshot algorithm {U. S. Department of Health and Human Services 2015} will be analyzed for the following subject subgroups (see Section 6.2.2.2 for details):

- Age (years): (a) < 50 and (b)  $\ge 50$
- Race: (a) black and (b) nonblack
- Region: (a) US and (b) Ex-US
- Study drug adherence (%): (a)  $\leq$  95 and (b)  $\geq$  95 (based on adherence up to Week 48 visit)

The proportion of subjects with hepatitis B virus (HBV) Deoxyribonucleic Acid (DNA) < 29 IU/mL at baseline and Week 48, and the change from baseline in log<sub>10</sub> HBV DNA by visit will be analyzed for the following subject subgroup:

• Subjects with HIV/HBV coinfection at baseline

#### 3.4.2. Subject Subgroups for Safety Analyses

Incidence of all treatment-emergent AEs (TEAEs) will be analyzed for the following subject subgroups:

- Age (years): (a)  $\leq 50$  and (b)  $\geq 50$
- Race: (a) black and (b) nonblack
- Region: (a) US and (b) Ex-US

Selected safety endpoints may be analyzed for the following subject subgroups (see Section 9.1 for details):

- Subjects with HIV/HBV coinfection at baseline
- Subjects with incident HIV/HBV coinfection while on study drug (if any)

Selected safety endpoints will be analyzed for the following subject subgroups (see Section 9.2 for details):

- Subjects with HIV/hepatitis C virus (HCV) coinfection at baseline
- Subjects with incident HIV/HCV coinfection while on study drug (if any)

Lastly, subgroup analysis by prior treatment regimen (ie, TDF-containing regimen versus non-TDF containing regimen) will be performed for the following endpoints:

- Urine retinal binding protein (RBP) to creatinine ratio
- beta-2 microglobulin to creatinine ratio
- Urine albumin to creatinine ratio (UACR)

## 3.5. Multiple Comparisons

The noninferiority evaluation of the proportion of subjects with HIV-1 RNA  $\geq$  50 copies/mL at Week 48 as determined by the US FDA-defined snapshot algorithm was the prespecified primary comparison. However, the Week 24 interim IDMC analysis was performed prior to the analysis for the primary endpoint and an alpha penalty of 0.00001 was applied for the Week 24 interim IDMC meeting. Therefore, the alpha level for the primary endpoint (ie, the proportion of subjects with HIV-1 RNA  $\geq$  50 copies/mL at Week 48 as determined by the US FDA-defined snapshot algorithm) was adjusted to 0.04999 (corresponding to 95.001% confidence interval [CI]) using both the FAS and the Week 48 PP analysis set. The alpha level for the key secondary efficacy endpoint, the proportion of subjects with HIV-1 RNA < 50 copies/mL at Week 48 as determined by the US FDA-defined snapshot algorithm, will also be adjusted to 0.04999 (corresponding to 95.001% CI) to be conservative using both the FAS and the Week 48 PP analysis set. No alpha level adjustment is applied other than for the primary and key secondary endpoints listed above.

### 3.6. Missing Data and Outliers

### 3.6.1. Missing Data

A missing datum for a given study analysis window may be due to any of the following reasons:

- A visit occurring in the window but data were not collected or were unusable
- A visit not occurring in the window
- A subject prematurely discontinuing from the study before reaching the window

In general, values for missing data will not be imputed, unless methods for handling missing data are specified.

For missing last dosing date of study drug, imputation rules are described in Section 3.8.1. The handling of missing or incomplete dates for AE onset is described in Section 7.1.5.2, and for concomitant non-antiretroviral (ARV) medications in Section 7.4.3.

#### **3.6.2. Outliers**

Outliers will be identified during the data management and data analysis process, but no sensitivity analyses will be done to evaluate the impact of outliers on efficacy or safety outcomes, unless specified otherwise. All data will be included in the analyses.

## 3.7. Data Handling Conventions and Transformations

Laboratory Data that are continuous in nature but are less than the lower limit of quantitation or above the upper limit of quantitation will be imputed as follows except for urine creatinine:

- A value that is 1 unit less than the limit of quantitation will be used for calculation of descriptive statistics if the datum is reported in the form of "< x" (where x is considered the limit of quantitation). For example, if the values are reported as < 50 and < 5.0, values of 49 and 4.9, respectively, will be used for calculation of summary statistics. An exception to this rule is any value reported as < 1 or < 0.1, etc. For values reported as < 1 or < 0.1, a value of 0.9 or 0.09, respectively, will be used for calculation of summary statistics.
- A value that is 1 unit above the limit of quantitation will be used for calculation of descriptive statistics if the datum is reported in the form of "> x" (where x is considered the limit of quantitation). Values with decimal points will follow the same logic as above.
- The limit of quantitation will be used for calculation of descriptive statistics if the datum is reported in the form of " $\leq$  x" or " $\geq$  x" (where x is considered the limit of quantitation).

For urine creatinine, a value of "< 1" is handled as a missing value in its summary and the calculation of related ratios.

Logarithm (base 10) transformation will be applied to HIV-1 RNA and HBV DNA data for efficacy analysis. HIV-1 RNA results of 'No HIV-1 RNA detected' and "<20 cp/mL HIV-1 RNA Detected" will be imputed as 19 copies/mL for analysis purpose. HBV DNA results of "<20 IU/mL HBV DNA detected" or "No HBV DNA detected" will be imputed as 19 IU/mL for analysis purpose. HCV RNA results of "<15 IU/mL HCV RNA detected" or "No HCV RNA detected" will be imputed as 14 IU/mL for analysis purpose.

Natural logarithm transformation will be used for analyzing concentrations in plasma samples. Concentration values that are below the lower limit of quantitation (BLQ) will be presented as "BLQ" in the concentration listing.

## 3.8. Analysis Windows

### 3.8.1. Definition of Study Day

**Study Day 1 (Randomized Phase)** is defined as the day when the first dose of the randomized study drug (ie, *B/F/TAF or SBR)* was taken, as recorded on the "Randomized Phase" Study Drug Administration eCRF.

**Study Day 1 (Extension Phase)** is defined as the day when the first dose of extension phase study drug (ie, *B/F/TAF*) was taken, as recorded on the "Extension Phase" Study Drug Administration eCRF. This day will only be available for subjects treated in the extension phase of the study.

**Study Days** are calculated relative to randomized phase Study Day 1. For events that occurred on or after the randomized phase Study Day 1, study days are calculated as (visit date minus randomized phase Study Day 1 plus 1). For events that occurred prior to the randomized phase Study Day 1, study days are calculated as (visit date minus randomized phase Study Day 1). All study days will be calculated from randomized phase Study Day 1 including observations collected from the extension phase of the study.

**Last Dose Date (Randomized Phase)** is defined as the latest of the randomized study drug end dates recorded on the "Randomized Phase" Study Drug Administration eCRF with "Permanently withdrawn" box checked for subjects who prematurely discontinued or completed the randomized study drug in the "Randomized Phase" according to the Study Drug Completion eCRF.

If the last dose date for randomized phase is missing (eg, only year of last dose date is known or completely missing due to lost to follow-up) for subjects who prematurely discontinued study drug or completed the study drug at the data cut date, the latest of nonmissing randomized study drug start dates and end dates, the clinical visit dates, and the laboratory visit dates, excluding the date of 30-day follow-up visit, from the randomized phase data, will be used to impute the randomized phase last dose date. For other partial missing last dose date, please see programming specification for imputation rule details. For subjects who are still on the randomized phase study drug, the data cut date will be used to impute the last dose date.

**Last Dose Date (Extension Phase)** is defined as the latest of the extension phase study drug end dates recorded on the "Extension Phase" Study Drug Administration eCRF with "Permanently Withdrawn" box checked for subjects who prematurely discontinued study drug according to the "Extension Phase" Study Drug Completion eCRF. This date will only be available for subjects treated in the extension phase of the study.

If the last dose date is missing for subjects who prematurely discontinued study drug in the extension phase of the study, the latest of nonmissing extension phase study drug start dates and end dates, the clinical visit dates, and the laboratory visit dates, excluding the date of 30-day follow-up visit, from the extension phase data, will be used to impute the extension phase last dose date. For subjects who are still on the extension phase study drug, the data cut date will be used to impute the last dose date.

Last Study Date is the latest of the randomized or extension phase (if available) study drug start dates and end dates, the clinic visit dates, and the laboratory visit dates, including the 30-day follow-up visit date, for subjects who prematurely discontinued study or who completed study according to the Study Completion eCRF. For subjects still on study, the last study date is defined to be the latest of data cut date, the clinic visit dates, and the laboratory visit dates, including the 30-day follow-up visit date. If subject died and the death date is complete (ie, not partial date) and before the imputed last study date, the complete death date should be used as the imputed last study date.

Baseline value is defined as the last value obtained on or prior to the randomized phase Study Day 1 for all assessments.

## 3.8.2. Analysis Windows

Subject visits might not occur on protocol specified days. Therefore, for the purpose of analysis, observations collected from the randomized phase of the study (ie, randomized phase data) will be assigned to analysis window. Observations collected from the extension phase of the study (ie, extension phase data) will not have analysis window assigned and will be included in listings with derived visit marked as "Extension". Any observations from the randomized phase in the "Post Week 48" window defined in Tables 3-2 to 3-5 will not be summarized in tables and figures, but included in listings.

The analysis windows for HIV-1 RNA, CD4+ cell count, CD4 %, HBV DNA, hematology, chemistry, urinalysis, urine pregnancy laboratory tests, eGFR<sub>CG</sub>, vital signs, and weight are presented in Table 3-2.

Table 3-2. Analysis Windows for HIV-1 RNA, CD4+ cell count, CD4 %, HBV DNA, Hematology, Chemistry, Urinalysis, and Urine Pregnancy Laboratory Tests, eGFR<sub>CG</sub>, Vital Signs, and Weight

| Visit ID | Nominal Day | Lower Limit | Upper Limit |
|--------------|-------------|-------------|-------------|
| Baseline | | | 1 |
| Week 4 | 28 | 2 | 42 |
| Week 8 | 56 | 43 | 70 |
| Week 12 | 84 | 71 | 126 |
| Week 24 | 168 | 127 | 210 |
| Week 36 | 252 | 211 | 294 |
| Week 48 | 336 | 295 | 378 |
| Post Week 48 | NA | 379 | |

Note: HBV DNA collection schedules are as follows: (1) For subjects who meet the definition of HBV infection at screening, HBV DNA will be collected at baseline, Weeks 4, 8, 12, 24, 36, and 48. (2) For subjects who meet the definition of HBV infection at any postbaseline visit, HBV DNA test will be performed at all subsequent visits. (3) For subjects who do not meet the definition of HBV infection at any visit, HBV DNA will be collected at baseline and Week 48.

The analysis windows for metabolic assessments (including fasting glucose and lipid panel: total cholesterol, high density lipoprotein [HDL], direct low density lipoprotein [LDL], triglycerides, and total cholesterol to HDL ratio) and HBV serology (including hepatitis B surface antibody [HBsAb], hepatitis B surface antigen [HBsAg], hepatitis B e-antigen [HBeAg], hepatitis B e-antibody [HBeAb], and hepatitis B core antibody [HBcAb]) are presented in Table 3-3.

Table 3-3. Analysis Windows for Metabolic Assessments and HBV Serology

| Visit ID | Nominal Day | Lower Limit | Upper Limit |
|--------------|-------------|-------------|-------------|
| Baseline | | | 1 |
| Week 12 | 84 | 2 | 126 |
| Week 24 | 168 | 127 | 252 |
| Week 48 | 336 | 253 | 420 |
| Post Week 48 | NA | 421 | |

Note: HBV serology collection schedules are as follows: (1) For subjects who meet the definition of HBV infection at screening, HBV serology will be collected at Weeks 12, 24, and Week 48. (2) For subjects who meet the definition of HBV infection at any postbaseline visit, HBV serology will be performed at all subsequent visits. (3) For subjects who do not meet the definition of HBV infection at any visit, HBV serology will be collected at baseline and Week 48.

The analysis windows for thyroid stimulating hormone (TSH; thyrotropin), renal function (including: urine albumin, urine creatinine, urine RBP, and urine beta-2 microglobulin, and derived ratios), and safety electrocardiogram (ECG) are presented in Table 3-4.

Table 3-4. Analysis Windows for TSH, Renal Function, and Safety ECG

| Visit ID | Nominal Day | Lower Limit | Upper Limit |
|--------------|-------------|-------------|-------------|
| Baseline | | | 1 |
| Week 24 | 168 | 2 | 252 |
| Week 48 | 336 | 253 | 420 |
| Post Week 48 | NA | 421 | |

The analysis windows for HCV serology and HCV RNA assessments are presented in Table 3-5.

Table 3-5. Analysis Windows for HCV Serology and HCV RNA Assessments

| Visit ID | Nominal Day | Lower Limit | Upper Limit |
|--------------|-------------|-------------|-------------|
| Baseline | | | 1 |
| Week 48 | 336 | 2 | 504 |
| Post Week 48 | NA | 505 | |

# 3.8.3. Selection of Data in the Event of Multiple Records in an Analysis Window

Depending on the statistical analysis method, single values are required for each analysis window. For example, change from baseline by visit usually requires a single value, whereas a time to event analysis would not require one value per analysis window. When a single value is needed, the following rule(s) will be used.

If multiple nonmissing numeric observations exist in a window, then records collected from the randomized phase of the study will be chosen as follows:

- For baseline, the latest available record on or prior to the first dose date of randomized study drug will be selected. If there are multiple records with the same collection time or no collection time recorded on the same day, average will be used for the baseline value, except for HIV-1 RNA (see below).
- For postbaseline visits:
  - For CD4+ cell count, CD4%, and HBV DNA, the record(s) collected on the latest day in the window will be selected for analysis.
  - For other numeric observations (eg, except HIV-1 RNA, CD4+ cell count, CD4%, and HBV DNA), the record(s) collected on the day closest to the nominal day for that visit will be selected. If there are 2 days equidistant from the nominal day, the later day will be selected.
  - For any numeric observations except HIV-1 RNA, if there are multiple records on the selected day, the arithmetic mean will be used.
- For baseline and postbaseline HIV-1 RNA, the latest (considering both collection date and time) record(s) in the window will be selected. If both "HIV RNA Taqman 2.0" and "HIV RNA Repeat" (ie, the HIV-1 RNA result obtained from an additional aliquot of the original sample) are available with the same collection time, the results from the "HIV RNA Repeat" will be selected for analysis purposes; otherwise, if there are multiple "HIV RNA Taqman 2.0" records with the same collection time, the geometric mean will be taken for analysis purposes.

If multiple valid nonmissing categorical observations exist in a window, records will be chosen as follows:

- For baseline, the last available record on or prior to the first dose date of randomized study drug will be selected. If there are multiple records with the same collection time or no collection time recorded on the same day, the value with the lowest severity will be selected (eg, normal will be selected over abnormal for safety ECG findings).
- For postbaseline visits, the most conservative value within the window will be selected (eg, abnormal will be selected over normal for safety ECG findings).

### 4. SUBJECT DISPOSITION

## 4.1. Subject Enrollment and Disposition

## 4.1.1. Subject Enrollment

The number and percentage of subjects randomized at each country, and investigator will be summarized by treatment group and overall using safety analysis set. The denominator for this calculation will be the number of subjects in the safety analysis set. Similarly, the number and percentage of subjects enrolled in each randomization stratum will be summarized using stratum assignment captured in the interactive web response system (IWRS).

If there are discrepancies between IWRS and ARV data with regard to stratum assignment, a listing of the discrepancies will be provided.

### 4.1.2. Subject Disposition

The summary of subject disposition will be provided by treatment group and overall for all screened subjects. This summary will include the number of subjects screened, screen failure subjects who were not randomized, subjects who met all eligibility criteria and were not randomized, subjects randomized but never treated, subjects in the safety analysis set, and subjects in FAS.

In addition, the number and percentage of the subjects in the following categories will be summarized:

- Still on study drug in the randomized phase, if applicable
- Completing study drug in the randomized phase
- Prematurely discontinuing study drug in the randomized phase (with summary of reasons for discontinuing study drug)
- Still on study in the randomized phase, if applicable
- Completing study in the randomized phase
- Prematurely discontinuing from study in the randomized phase (with summary of reasons for discontinuing study)
- Entering and treated in the extension phase
- Subjects still on study drug in the extension phase
- Prematurely discontinuing study drug in the extension phase

The denominator for the percentages of subjects in each category, except for the categories of "subjects still on study drug in the extension phase" and "prematurely discontinuing study drug in the extension phase", will be the number of subjects in the safety analysis set. The denominator for the percentage of subjects in the categories of "subjects still on study drug in the extension phase" and "prematurely discontinuing study drug in the extension phase" will be the numbers of subjects entering and treated in the extension phase.

No inferential statistics will be generated. A data listing of reasons for premature study drug/study discontinuation will be provided.

### 4.2. Extent of Study Drug Exposure and Adherence

### 4.2.1. Duration of Exposure to Randomized Study Drug

Duration of exposure to randomized study drug is defined as (the randomized phase last dose date – the randomized phase first dose date + 1), regardless of temporary interruptions in study drug administration, and will be expressed in weeks using up to 1 decimal place (eg, 4.5 weeks). For the calculation of the duration of exposure to study drug, the data cut date will be used to impute the last dose date for subjects who have not permanently discontinued the randomized phase of the study at the time of the data cut date.

Duration of exposure to randomized study drug will be summarized using descriptive statistics (n, mean, SD, median, Q1, Q3, minimum, and maximum) and as the number and percentage of subjects exposed for specified periods, eg,  $\geq$  4 weeks (28 days),  $\geq$  8 weeks (56 days),  $\geq$  12 weeks (84 days),  $\geq$  24 weeks (168 days),  $\geq$  36 weeks (252 days),  $\geq$  48 weeks (336 days), etc.

Summaries will be provided by treatment group for subjects in the safety analysis set. No inferential statistics will be provided.

Time to premature discontinuation of randomized study drug will be analyzed using the Kaplan-Meier (KM) method by treatment group based on the safety analysis set. The log rank test will be used to compare the difference in study drug exposure between the 2 randomized treatment groups. Subjects who completed 48-week randomized phase of the study treatment will be censored at the last dose date of the randomized study drug. Subjects who are still on the randomized study drug will be censored at the imputed last dose date (ie, data cut date). A plot of KM estimates for the time to premature discontinuation of the randomized study drug by treatment group will be generated.

## 4.2.2. Adherence to Study Drug Regimen

Study drug regimen adherence will be computed based on pill counts of each randomized study drug included in that study drug regimen. The numbers of pills of randomized phase study drug (ie, B/F/TAF, GEN, STB, ATV, RTV, or FTC/TDF) dispensed and returned are captured on study drug accountability eCRF.

Adherence (%) of a study drug regimen (Note: study drug regimen only includes 1 study drug for B/F/TAF, GEN, STB, and 3 study drugs for ATV+RTV+FTC/TDF) will be calculated as follows for pills dispensed in the randomized phase of the study:

Adherence (%) = 
$$100 \times \frac{\text{Total No. of pills taken}}{\text{Total No. of pills prescribed}}$$
  
=  $100 \times \frac{\sum \sum \text{No. of pills taken at each dispensing period for each drug}^{[1]}}{\sum \sum \text{No. of pills prescribed at each dispensing period for each drug}^{[2]}}$ 

- [1] Number of pills taken at a distinct dispensing period for a study drug is calculated as the minimum of (a) the daily number of pills prescribed for the study drug multiplied by the duration of treatment at the dispensing period of the same dispensing date, and (b) the number of pills taken for the study drug (number of pills dispensed minus the number of pills returned). Total number of pills taken is determined by summing the number of pills taken for each study drug contained in the study drug regimen from all evaluable dispensing periods.
- [2] Number of pills prescribed at a distinct dispensing period for a study drug is calculated as the daily number of pills prescribed for the study drug multiplied by the duration of treatment at the dispensing period of the same dispensing date. Total number of pills prescribed is determined by summing the number of pills prescribed for each study drug contained in the study drug regimen from all evaluable dispensing periods.

The duration of treatment at a dispensing period for a study drug is calculated as the minimum of (a) the last returned date of the same dispensing period for the study drug, (b) date of premature discontinuation of the study drug, and (c) <u>next pill dispensing date</u> of the study drug, minus dispensing date of the study drug.

The next pill dispensing date is the following dispensing date of the study drug regardless of the bottle return date.

For a record where the number of pills returned was missing (with "Yes" answered for "Was Bottle returned?" question), it is assumed the number of pills returned was zero. If the number of pills dispensed was missing or any study drug bottle was not returned or the bottle return status was unknown, all records in that dispensing period for that study drug will be excluded from both denominator and numerator calculation.

Adherence up to Week 48 visit (ie, overall adherence for the randomized phase of the study) will be calculated using all data from the entire dosing period up to the date of permanent discontinuation of the randomized study drugs.

Descriptive statistics for adherence up to Week 48 visit for a study drug regimen (n, mean, SD, median, Q1, Q3, minimum, and maximum) along with the number and percentage of subjects belonging to adherence categories (eg,  $< 80\%, \ge 80\%$  to  $< 90\%, \ge 90\%$  to  $< 95\%, \ge 95\%$ ) will be provided by treatment group for subjects who return at least 1 bottle and have calculable adherence during the randomized phase of the study in the safety analysis set. No inferential statistics will be provided.

## 4.3. Protocol Deviations

A listing will be provided for all randomized subjects who violated at least 1 inclusion or exclusion criterion. The listing will include the criteria not met. A listing of subjects who received the wrong study drug will also be provided.

### 5. BASELINE CHARACTERISTICS

## **5.1.** Demographics and Baseline Characteristics

Subject demographic data (eg, age, sex at birth, race, and ethnicity) and baseline characteristics (eg, body weight, height, and body mass index [BMI]) will be summarized by treatment group and overall using descriptive statistics (n, mean, SD, median, Q1, Q3, minimum, and maximum) for continuous data and by the number and percentage of subjects for categorical data. The summaries of demographic data and baseline characteristics will be provided for the safety analysis set.

For categorical data, the Cochran-Mantel-Haenszel (CMH) test (ie, general association statistic for nominal data) will be used to compare the 2 treatment groups. For continuous data, the 2-sided Wilcoxon rank sum test will be used to compare the 2 treatment groups.

### **5.2.** Baseline Disease Characteristics

The following baseline disease characteristics will be summarized:

- HIV-1 RNA categories (copies/mL): (a)  $\leq 50$ , (b)  $\geq 50$
- CD4+ cell count (/μL)
- CD4+ cell count categories (/ $\mu$ L): (a) < 50, (b)  $\geq$  50 to < 200, (c)  $\geq$  200 to < 350, (d)  $\geq$  350 to < 500, and (e)  $\geq$  500
- CD4 percentage (%)
- Mode of infection (HIV risk factors)
- HIV disease status
- eGFR<sub>CG</sub> (mL/min )
- Medical history: diabetes mellitus (Yes/No), hypertension (Yes/No), cardiovascular disease (Yes/No), and hyperlipidemia (Yes/No) (see Appendix 3 for details)
- HIV/HBV coinfection status (Yes/No/Missing, see Section 9.1 for definition)
- HIV/HCV coinfection status (Yes/No/Missing, see Section 9.2 for definition)
- Smoking status: (a) Never Smoker, (b) Former Smoker, and (c) Current Smoker (see Appendix 5 for details)
- Prior ARV regimen: (a) E/C/F/TAF, (b) E/C/F/TDF; (c) RTV boosted ATV + FTC/TDF (see Section 7.4.2 and Appendix 5 for details)

For categorical data, the Cochran-Mantel-Haenszel (CMH) test (general association statistic for nominal data, and row means scores differ statistic for ordinal data) will be used to compare the 2 treatment groups. For continuous data, the 2-sided Wilcoxon rank sum test will be used to compare the 2 treatment groups.

## **5.3.** Medical History

General medical history data will be collected at screening and listed only. General medical history data will be coded using the current version of Medical Dictionary for Regulatory Activities (MedDRA).

### 6. EFFICACY ANALYSES

### 6.1. Primary Efficacy Endpoint

## 6.1.1. Definition of the Primary Efficacy Endpoint

The primary efficacy endpoint is the proportion of subjects with HIV-1 RNA  $\geq$  50 copies/mL at Week 48 as determined by the US FDA-defined snapshot algorithm {U. S. Department of Health and Human Services 2015}. The proportions are expressed as percentages for presentation purposes.

## 6.1.2. US FDA-defined Snapshot Algorithm

The analysis window at Week 48 is defined as from Study Day 295 to Study Day 378, inclusive. All HIV-1 RNA data collected on-treatment (ie, data collected up to 1 day after the randomized phase last dose date) will be used in the US FDA-defined snapshot algorithm. Virologic outcome will be defined as the following categories:

- **HIV-1 RNA < 50 copies/mL:** this includes subjects who have the last available on-treatment HIV-1 RNA < 50 copies/mL in the Week 48 analysis window
- HIV-1 RNA  $\geq$  50 copies/mL: this includes subjects
  - a. Who have the last available on-treatment HIV-1 RNA ≥ 50 copies/mL in the Week 48 analysis window, or
  - b. Who do not have on-treatment HIV-1 RNA data in the Week 48 analysis window and
    - 1) Who discontinue study drug prior to or in the Week 48 analysis window due to lack of efficacy, or
    - 2) Who discontinue study drug prior to or in the Week 48 analysis window due to AE or death and have the last available on-treatment HIV-1 RNA  $\geq$  50 copies/mL, or
    - 3) Who discontinue study drug prior to or in the Week 48 analysis window due to reasons other than AE, death, or lack of efficacy and have the last available on-treatment HIV-1 RNA ≥ 50 copies/mL
- No Virologic Data in the Week 48 Window: this includes subjects who do not have ontreatment HIV-1 RNA data in the Week 48 analysis window because of the following:
  - a. Discontinuation of study drug prior to or in the Week 48 analysis window due to AE or death and the last available on-treatment HIV-1 RNA < 50 copies/mL, or

- b. Discontinuation of study drug prior to or in the Week 48 analysis window due to reasons other than AE, death, or lack of efficacy and the last available on-treatment HIV-1 RNA < 50 copies/mL or,
- c. Missing data during the window but on study drug.

The flowchart of the US FDA-defined snapshot algorithm is provided in Appendix 2.

The Week 48 virologic outcomes for the US FDA-defined snapshot algorithm will be listed.

Note: For switch trials, the US FDA-defined snapshot algorithm classifies subjects who discontinue study drug due to AE or death and have the last available on-treatment HIV-1 RNA value  $\geq 50$  copies/mL in the "HIV-1 RNA  $\geq 50$  copies/mL" category. For treatment naive study population, these subjects will be classified in the "No Virologic Data in the Week 48 Window" category.

## 6.1.3. Statistical Hypothesis for the Primary Efficacy Endpoint

**Null hypothesis**: the B/F/TAF group (Treatment Group 1) is at least 4% higher than the SBR group (Treatment Group 2) with respect to the proportion of subjects with HIV-1 RNA ≥ 50 copies/mL as determined by the US FDA-defined snapshot algorithm at Week 48.

**Alternative hypothesis**: the B/F/TAF group (Treatment Group 1) is less than 4% higher than the SBR group (Treatment Group 2) with respect to the proportion of subjects with HIV-1 RNA ≥ 50 copies/mL at Week 48.

### 6.1.4. Primary Analysis of the Primary Efficacy Endpoint

The analysis purpose of the primary efficacy endpoint is to assess the noninferiority of switching to B/F/TAF relative to continuing on SBR. Noninferiority will be assessed using a conventional 95% CI approach, with a noninferiority margin of 4%.

For the interim analysis performed for the IDMC at Week 24, an alpha of 0.00001 has been spent. Therefore, the significance level for the 2-sided test in the primary analysis at Week 48 will be 0.04999 (corresponding to 95.001% CI).

The point estimate of treatment difference (B/F/TAF group – SBR group) in the percentage of subjects with HIV-1 RNA  $\geq$  50 copies/mL and the associated 2-sided 95.001% CI will be constructed based on an unconditional exact method using 2 inverted 1-sided tests.

It will be concluded that B/F/TAF is noninferior to SBR if the upper bound of the 2-sided 95.001% CI of the difference (B/F/TAF group – SBR group) in the percentage of subjects with HIV-1 RNA  $\geq$  50 copies/mL is less than 4%.

The number and percentage of subjects with HIV-1 RNA < 50 copies/mL, HIV-1 RNA ≥ 50 copies/mL, and reasons for no virologic data at Week 48 will be summarized.

If noninferiority of B/F/TAF versus SBR is established, the same 95.001% CI used in evaluating noninferiority at Week 48 will be used to evaluate superiority. If the upper bound of the 95.001% CI is less than 0, superiority of B/F/TAF over SBR is established. The 2-sided Fisher's exact test will also be used to assess superiority as a secondary assessment.

The FAS will be used for the primary efficacy endpoint analysis and the superiority evaluation.

### 6.1.5. Secondary Analysis of the Primary Efficacy Endpoint

A secondary analysis based on the Week 48 PP analysis set will also be performed to evaluate the robustness of the primary analysis of the primary endpoint. For this secondary analysis, 95.001% CI for the treatment difference in the primary efficacy endpoint will also be evaluated based on an unconditional exact method using 2 inverted 1-sided tests.

### **6.2.** Secondary Efficacy Endpoints

## 6.2.1. Definition of the Secondary Efficacy Endpoints

The secondary efficacy endpoints include:

- The proportion of subjects with HIV-1 RNA < 50 copies/mL at Week 48 as determined by the US FDA-defined snapshot algorithm
- The change from baseline in CD4+ cell count at Week 48

## 6.2.2. Analysis of the Secondary Efficacy Endpoints

6.2.2.1. Analysis of the Proportion of Subjects with HIV-1 RNA < 50 copies/mL as Determined by US FDA-defined Snapshot Algorithm

The proportion of subjects with HIV-1 RNA < 50 copies/mL at Week 48 as determined by the US FDA-defined snapshot algorithm will be analyzed similarly to the primary efficacy endpoint. However, the noninferiority margin used for this endpoint will be 10%.

Similarly to the primary efficacy endpoint, noninferiority will be assessed using the conventional CI approach. The point estimate of treatment difference (B/F/TAF group – SBR group) in the percentage of subjects with HIV-1 RNA < 50 copies/mL and the associated 2-sided 95.001% CI will be constructed based on an unconditional exact method using 2 inverted 1-sided tests.

It will be concluded that B/F/TAF is noninferior to SBR if the lower bound of the 2-sided 95.001% CI of the difference between treatment groups (B/F/TAF group – SBR group) in the percentage of subjects with HIV-1 RNA < 50 copies/mL is greater than -10%.

The above analysis will be performed using both the FAS and the Week 48 PP analysis set.

In addition, the following analyses will be performed using the FAS to evaluate the interaction between country and treatment to assess homogeneity of treatment effect across different countries.

For each country, the difference in the proportion of subjects with HIV-1 RNA < 50 copies/mL between treatment groups and its 95% CI will be calculated based on an unconditional exact method using 2 inverted 1-sided tests.

The CMH analysis will be used to estimate the odds ratio and corresponding 95% CI for each country and overall. The homogeneity of the odds ratios across different countries will be tested using a Breslow-Day test and a corresponding p-value will be reported.

6.2.2.2. Subgroup Analysis of the Proportion of Subjects with HIV-1 RNA < 50 copies/mL as Determined by US FDA-defined Snapshot Algorithm

The proportion of subjects with HIV-1 RNA  $\geq$  50 copies/mL at Week 48 as determined by the US FDA-defined snapshot algorithm (primary endpoint) is expected to be very low (around 2%). The efficacy analysis by subgroup will be conducted by assessing the proportion of subjects with HIV-1 RNA < 50 copies/mL, determined by the US FDA-defined snapshot algorithm at Week 48 (a secondary efficacy endpoint) within each subgroup specified in Section 3.4.1 based on the FAS.

For each level of subgroup factors, the proportion difference between treatment groups and the associated 2-sided 95% CIs will be computed based on an unconditional exact method using 2 inverted 1-sided tests.

Additionally, a logistic regression model will be performed which include subgroup factor, treatment, and treatment by subgroup factor. The odds ratio and the associated 95% CI will be estimated within each subgroup. The homogeneity of the treatment effects between subgroups will be evaluated using a Wald test based on the interaction between treatment and the subgroup factor.

A forest plot of the treatment differences in HIV-1 RNA < 50 copies/mL (US FDA-defined snapshot algorithm) at Week 48 and their associated 95% CIs for each subgroup will be generated.

### 6.2.2.3. Analysis of CD4+ Cell Count

All CD4+ cell count will be summarized using observed, on-treatment data (ie, data collected up to 1 day after the randomized phase last dose date) for subjects in the FAS and in the Week 48 PP analysis set, respectively.

The changes from baseline in CD4+ cell count at Week 48 will be summarized by treatment group using descriptive statistics. The differences in changes from baseline in CD4+ cell count between the 2 treatment groups and the associated 95% CI will be constructed using analysis of variance (ANOVA) models, including treatment group as a fixed effect. The change from baseline in CD4+ cell count will also be summarized at visits other than Week 48 by treatment group.

The mean and 95% CI of change from baseline in CD4+ cell count over time will be plotted for the FAS.

In addition, the change from baseline in CD4+ cell counts with missing values imputed using the last observation carried forward (LOCF) method will be summarized at each visit based on the FAS. The algorithm for LOCF is as follows:

- If a value is missing in an analysis visit window, the missing value will be replaced with the
  last on-treatment value (ie, data collected up to 1 day after the randomized phase last dose
  date) observed before the analysis visit window that has the missing value.
- Baseline values will be carried forward to impute the postbaseline value at a specific visit, if there is no nonmissing postbaseline observation collected prior to that visit.

## 6.3. Tertiary Efficacy Endpoints

## 6.3.1. Definition of the Tertiary Efficacy Endpoints





# 6.4. Changes From Protocol-Specified Efficacy Analyses

No change from protocol-specified efficacy analysis is planned.

### 7. SAFETY ANALYSES

Safety data from the randomized phase of the study (ie, randomized phase data) will be summarized for the subjects in the safety analysis set. All safety data collected up to 30 days after the randomized phase last dose date will be summarized by treatment group, unless specified otherwise. All safety data from both phases of the study will be included in data listings.

#### 7.1. Adverse Events and Deaths

## 7.1.1. Adverse Event Dictionary

Clinical and laboratory AEs will be coded using the current version of MedDRA. System organ class (SOC), high-level group term (HLGT), high-level term (HLT), preferred term (PT), and lower-level term (LLT) will be provided in the AE dataset.

## **7.1.2.** Adverse Event Severity

Adverse events are graded by the investigator as Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe) or Grade 4 (life threatening) according to toxicity criteria specified in the protocol. The severity grade of events for which the investigator did not record severity will be left as "missing" data listings.

# 7.1.3. Relationship of Adverse Events to Study Drug

Related AEs are those for which the investigator selected "Related" on the AE eCRF to the question of "Related to Study Treatment." Events for which the investigator did not record relationship to study drug will be considered related to study drug for summary purposes. However, by-subject data listings will show the relationship as missing.

#### 7.1.4. Serious Adverse Events

Serious adverse events (SAEs) will be identified and captured as SAEs if AEs met the definitions of SAE specified in the study protocol. Serious adverse events captured and stored in the clinical database will be reconciled with the SAE database from the Gilead Drug Safety and Public Health (DSPH) Department before data finalization.

### 7.1.5. Treatment-Emergent Adverse Events

### 7.1.5.1. Definition of Treatment-Emergent Adverse Events

Treatment-emergent adverse events (TEAEs) are defined as 1 or both of the following:

- Any AEs with an onset date on or after the study drug start date and no later than 30 days after permanent discontinuation of the study drug, or
- Any AEs leading to premature discontinuation of study drug

The TEAE definitions will be applied to the randomized phase data and the extension phase data, separately. When randomized phase data are used, AEs onset date will be compared with the randomized phase first dose date and last dose date and premature discontinuation of study drug refers to study drug discontinuation in the randomized phase. An AE meeting the TEAE criteria will be considered as a TEAE in the randomized phase. When extension phase data are used, AEs onset date will be compared with the extension phase first dose date and last dose date and premature discontinuation of study drug refers to study drug discontinuation in the extension phase. An AE meeting the TEAE criteria will be considered as a TEAE in the extension phase.

## 7.1.5.2. Incomplete Dates

If the onset date of the AE is incomplete and the AE stop date is not prior to the first dosing date of randomized study drug, the month and year (or year alone if month is not recorded) of onset determine whether an AE is treatment emergent.

The event is considered treatment emergent for the randomized phase if both of the following 2 criteria are met:

- The month and year (or year) of the AE onset is **the same as or after** the month and year (or year) of the first dosing date of randomized study drug, and
- The month and year (or year) of the AE onset is **the same as or before** the month and year (or year) of the date corresponding to the minimum of (1) the randomized phase last dose date plus 30 days AND (2) the extension phase first dose date minus 1 day

The event is considered treatment emergent for the extension phase if both of the following 2 criteria are met:

- The month and year (or year) of the AE onset is **after** the month and year (or year) of the first dosing date of extension phase study drug, and
- The month and year (or year) of the AE onset is **the same as or before** the month and year (or year) of the date corresponding to 30 days after the date of the last dose of extension phase study drug

An AE with completely missing onset and stop dates, or with the onset date missing and a stop date marked as ongoing or on or after the first dosing date of randomized study drug, will be considered as a TEAE for the randomized phase. In addition, an AE with the onset date missing and incomplete stop date with the same or later month and year (or year alone if month is not recorded) as the first dosing date of the randomized study drug will be considered as a TEAE for the randomized phase.
## 7.1.6. Summaries of Adverse Events and Death

Only TEAEs in the randomized phase will be included in the summary tables. The number and percentage of subjects who experienced at least 1 TEAE will be provided and summarized by SOC, HLT, PT, and treatment group. For other AEs reported in the randomized phase and described below, summaries will be provided by SOC, PT, and treatment group using the safety analysis set:

- Any Grade 2, 3, or 4 treatment-emergent AEs
- Any Grade 3 or 4 treatment-emergent AEs
- All treatment-emergent study drug-related AEs
- Any Grade 2, 3, or 4 treatment-emergent study drug-related AEs
- Any Grade 3 or 4 treatment-emergent study drug-related AEs
- All treatment-emergent SAEs
- All treatment-emergent study drug-related SAEs
- All treatment-emergent AEs that caused premature discontinuation from study drug

A brief, high-level summary of AEs described above will be provided by treatment group and by the number and percentage of subjects who experienced the above AEs. Treatment-emergent deaths observed in the randomized phase will be also included in this summary.

Treatment-emergent death refers to deaths that occurred between the randomized phase first dose date and the randomized phase last dose date plus 30 days (inclusive).

Multiple events will be counted only once per subject in each summary. Adverse events will be summarized and listed first in alphabetic order of SOC and HLT within each SOC (if applicable), and then by PT in descending order of total frequency within each SOC. For summaries by severity grade, the most severe grade will be used for those AEs that occurred more than once in an individual subject during the study.

In addition to the above summary tables, all TEAEs, Grade 3 or 4 TEAEs, treatment-emergent study drug-related AEs, Grade 2, 3, or 4 treatment-emergent study drug-related AEs, and treatment-emergent SAEs will be summarized by PT only, in descending order of total frequency.

In addition, data listings for all AEs regardless of the study phases will be provided for the following:

- All AEs
- Grade 3 and 4 AEs

- SAEs
- Study-Drug-Related SAEs
- Deaths report
- AEs leading to premature discontinuation of study drug

## 7.1.7. Additional Analysis of Adverse Events

## 7.1.7.1. Stage 3 Opportunistic Illnesses in HIV

On an ongoing basis, AEs will be reviewed for events that might meet the definition of stage 3 opportunistic illnesses in HIV that are indicative of an AIDS-defining diagnoses (see Protocol Appendix 5). The Gilead medical monitor will review the possible stage 3 opportunistic illnesses and approve the events that meet the definition. Events that meet the stage 3 opportunistic illness definition of an AIDS-defining diagnosis will be listed.

#### 7.1.7.2. Cardiovascular or Cerebrovascular Events

Preferred terms for defining cardiovascular or cerebrovascular events are from relevant Standardised MedDRA Query (SMQ). The selected PT listing was provided by Gilead DSPH and reviewed by Gilead medical monitors, which is the same PT listing used to search "Cardiovascular Disease" medical history (see details in Appendix 3).

The number and percentage of subjects with treatment-emergent cardiovascular or cerebrovascular events and serious cardiovascular or cerebrovascular events by PT will be provided by treatment group based on the safety analysis set. Statistical comparisons of the subject incidence rates between the 2 treatment groups will be performed using the Fisher's exact test. A data listing of cardiovascular or cerebrovascular events will be provided.

## 7.1.7.3. Hepatic Events

Preferred terms for defining hepatic events are from 15 relevant SMQs, which are identified as non-infectious and non-congenital hepatobiliary disorders. The selected PT listing was provided by Gilead DSPH and reviewed by Gilead medical monitors (see details in Appendix 4).

The number and percentage of subjects with treatment-emergent hepatic events and serious hepatic events by PT will be summarized by treatment group based on the safety analysis set. Statistical comparisons of the subject incidence rates between the 2 treatment groups will be performed using Fisher's exact test. A data listing of hepatic events will be provided.

## 7.2. Laboratory Evaluations

Laboratory data collected during the randomized phase of the study will be analyzed and summarized using both quantitative and qualitative methods. Summaries of laboratory data will be provided for the safety analysis set. The analysis will be based on values reported in conventional units. When values are below the LOQ, they will be listed as such, and the imputed value will be used for the purpose of calculating summary statistics as specified in Section 3.7.

A by-subject listing for laboratory test results will be provided by subject ID number and visit in chronological order for hematology, serum chemistry, and urinalysis separately for all data collected from both phases of the study. Values falling outside of the reference range and/or having a severity grade of 1 or higher on the Gilead Grading Scale for Severity of Adverse Events and Laboratory Abnormalities will be flagged in the data listings, as appropriate.

## 7.2.1. Summaries of Numeric Laboratory Results

Descriptive statistics will be provided by treatment group for each laboratory test specified in the study protocol as follows:

- Baseline values
- Values at each postbaseline analysis window
- Change from baseline at each postbaseline analysis window
- Percentage change from baseline to each postbaseline analysis window (if specified)

A baseline laboratory value will be defined as the last nonmissing value obtained on or prior to the date of first dose of randomized study drug. Change from baseline to a postbaseline visit will be defined as the postbaseline value minus the baseline value. The mean, median, Q1, Q3, minimum, and maximum values will be displayed to the reported number of digits; SD values will be displayed to the reported number of digits plus 1.

In the case of multiple values in an analysis window, data will be selected for analysis as described in Section 3.8.3.

#### **Calcium Corrected for Albumin**

Calcium corrected for albumin will be calculated and summarized for the study. The following formula will be used when both serum calcium and albumin results for a given blood drawn are available and serum albumin value is < 4.0 g/dL.

Calcium corrected for albumin (mg/dL) = serum calcium (mg/dL) + 0.8 x (4.0 – albumin (g/dL)).

Toxicity grading for calcium will be applied based on the corrected values.

## **Estimate GFR**

The following formulae will be used to calculate eGFR<sub>CG</sub>:

• eGFR(CG) (mL/min) =  $[(140 - age (yrs)) \times weight (kg) \times (0.85 if female)] / (SCr (mg/dL) \times 72)$ , where weight is total body mass in kilograms.

## 7.2.2. Graded Laboratory Values

The Gilead Grading Scale for Severity of Adverse Events and Laboratory Abnormalities will be used for assigning toxicity grades (0 to 4) to laboratory results for analysis. Grade 0 includes all values that do not meet the criteria for an abnormality of at least Grade 1. For laboratory tests with criteria for both increased and decreased levels, analyses for each direction (ie, increased, decreased) will be presented separately.

If there is any laboratory toxicity grading scale overlapping with the normal reference ranges (eg, grade 1 scale overlaps with normal reference ranges), laboratory values that are within the normal range will be grade 0, except for lipid tests.

For triglycerides, LDL, and cholesterol, protocol-specified toxicity grading scale is for fasting test values, so nonfasting lipid results (or lipid results without a known fasting status) will not be graded or summarized by toxicity grades.

For the international normalized ratio (INR) of prothrombin time (PT), protocol-specified toxicity grading scale depends on the upper limit of normal range (ULN). While the ULN of INR depends on whether the subject is taking anticoagulant medication or not (ie, Not taking oral anticoagulant: 0.8 - 1.2; Taking oral anticoagulant: 2.0 - 3.0), this information is not collected by the reference laboratory. As a result, INR will be graded by assuming subject is not taking an oral anticoagulant, which is a conservative approach that may lead to over-reporting of abnormalities for INR. Consequently, INR and PT will not be included in summaries of laboratory abnormalities, but will be included in listings for the following reasons: 1) INR and PT are reflexive tests; 2) only the absolute values, not the toxicity grade, are needed for subject management purposes; and 3) more importantly, the toxicity grades for INR may be over-reported.

## 7.2.2.1. Treatment Emergent Laboratory Abnormalities

Treatment-emergent laboratory abnormalities are defined as values that increase at least 1 toxicity grade from baseline at any postbaseline time point, up to 30 days from the randomized phase last dose date. If the relevant baseline laboratory value is missing, any abnormality of at least Grade 1 observed within the time frame specified above will be considered treatment-emergent.

Fasting glucose and nonfasting glucose (including glucose results without a known fasting status) are graded based on different grading scales as specified in the protocol.

Treatment-emergent laboratory abnormalities will be summarized for fasting glucose. Maximum postbaseline grade, instead of treatment-emergent grade, for nonfasting glucose (including glucose results without a known fasting status) will be summarized, as nonfasting glucose was not assessed at baseline visit for most of the subjects; therefore, an abnormality is treatment-emergent or not cannot be determined for these subjects.

Both urine RBC based on microscopic examination, labeled as Hematuria (Quantitative), and urine blood based on dipstick, labeled as Hematuria (Dipstick), are assessed routinely and assigned a toxicity grade in this study. Urine RBC based on microscopic examination will be presented in laboratory toxicity summary tables and listings while urine blood based on dipstick will be presented in the listings only.

## 7.2.2.2. Summaries of Laboratory Abnormalities

The following summaries (number and percentage of subjects) for treatment-emergent laboratory abnormalities will be provided by lab test and treatment group; subjects will be categorized according to the most severe postbaseline abnormality grade for a given lab test:

- Treatment-emergent laboratory abnormalities
- Treatment-emergent Grade 3 and 4 laboratory abnormalities
- Treatment-emergent Grade 2, 3, and 4 laboratory abnormalities

For all summaries of laboratory abnormalities, the denominator is the number of subjects with any nonmissing postbaseline values up to 30 days after the randomized phase last dose date.

A by-subject listing of all treatment-emergent laboratory abnormalities and treatment-emergent Grade 3 or 4 laboratory abnormalities will be provided by subject ID number and visit in chronological order.

## 7.2.3. Metabolic Laboratory Evaluations

For metabolite assessments, including fasting glucose and the lipid panel (ie, total cholesterol, triglycerides, LDL, HDL, total cholesterol to HDL ratio), only those measurements under fasting status will be summarized. P-values comparing the difference between the 2 treatment groups in baseline values and the change from baseline in metabolic assessment will be estimated from the 2-sided Wilcoxon rank sum test.

In addition, the number and percentage of subjects who took lipid modifying medications at study entry and initiated the medications during the randomized phase of the study will be provided, respectively. Statistical comparisons of the subject incidence rates between the 2 treatment groups will be performed using Fisher's exact test.

A lipid modifying medication is defined as a medication with drug class = "LIPID MODIFYING AGENTS" and CMDECOD containing the wording of "STATIN".

A sensitivity analysis of fasting lipid tests will be performed by excluding subjects who took lipid modifying medications at study entry or initiated the medications during the randomized phase of the study: baseline values, Week 48 values, and changes from baseline at Week 48 will be summarized by treatment group using descriptive statistics. Baseline and change from baseline at Week 48 will be compared between the 2 treatment groups using a 2-sided Wilcoxon rank sum test. Only subjects with both baseline and Week 48 postbaseline values will be included in the analysis.

Median (Q1, Q3) of change from baseline in fasting metabolic assessments over time will be plotted by treatment group.

## 7.2.4. Liver-Related Laboratory Evaluations

Liver-related abnormalities after initial study drug dosing will be examined and summarized using the number and percentage of subjects who were reported to have the following laboratory test values for postbaseline measurements collected in the randomized phase of this study:

- Aspartate aminotransferase (AST): (a) > 3 × ULN, (b) > 5 × ULN, (c) > 10 × ULN,
  (d) > 20 × ULN
- Alanine aminotransferase (ALT): (a) > 3 × ULN, (b) > 5 × ULN, (c) > 10 × ULN,
  (d) > 20 × ULN
- AST or ALT: (a)  $> 3 \times ULN$ , (b)  $> 5 \times ULN$ , (c)  $> 10 \times ULN$ , (d)  $> 20 \times ULN$
- Total bilirubin: (a)  $> 1 \times ULN$ , (b)  $> 2 \times ULN$
- Alkaline phosphatase (ALP)  $> 1.5 \times ULN$
- AST or ALT >  $3 \times ULN$  and total bilirubin: (a) >  $1.5 \times ULN$ , (b) >  $2 \times ULN$
- AST or ALT  $> 3 \times ULN$  and total bilirubin  $> 2 \times ULN$  and ALP  $< 2 \times ULN$

The summary will include data from all postbaseline visits up to 30 days after the randomized phase last dose date. For individual laboratory tests, subjects will be counted once based on the most severe postbaseline value. For both the composite endpoint of AST or ALT and total bilirubin, and the composite endpoint of AST or ALT, total bilirubin, and ALP, subjects will be counted once when the criteria are met at the same postbaseline visit date. The denominator is the number of subjects in the safety analysis set with nonmissing postbaseline value of the tests in evaluation at the same postbaseline visit date.

Subjects with AST or ALT  $> 3 \times ULN$  will also be listed.

In addition, baseline, postbaseline, and change from baseline in AST, ALT, ALP, and total bilirubin will be summarized by treatment group and visit using descriptive statistics. Baseline and change from baseline will be compared between the 2 treatment groups using a 2-sided Wilcoxon rank sum test

Furthermore, ALT flare, defined as subjects with ALT elevation > 2 x Baseline ALT and > 10 x ULN and confirmed at 2 consecutive visits, will be evaluated and listed for subjects with HIV/HBV coinfection at baseline.

## 7.2.5. Renal-Related Laboratory Evaluations

### 7.2.5.1. Serum Creatinine and eGFR<sub>CG</sub>

Baseline, postbaseline, and change from baseline in serum creatinine and  $eGFR_{CG}$  will be summarized by treatment group and visit using descriptive statistics. Baseline and change from baseline will be compared between the 2 treatment groups using a 2-sided Wilcoxon rank sum test.

Median (Q1, Q3) of change from baseline in serum creatinine and eGFR<sub>CG</sub> over time will be plotted by treatment group.

7.2.5.2. Urine Creatinine, Urine Retinol Binding Protein to Creatinine Ratio, and Beta-2-Microglobulin to Creatinine Ratio

Baseline, postbaseline, change from baseline, and percentage change from baseline in urine RBP to creatinine ratio and beta-2 microglobulin to creatinine ratio will be summarized by treatment group and visit using descriptive statistics. Baseline and percentage change from baseline will be compared between the 2 treatment groups using a 2-sided Wilcoxon rank sum test.

Median (Q1, Q3) percentage change from baseline in urine RBP to creatinine ratio and beta-2 microglobulin to creatinine ratio over time will be plotted by treatment group.

Baseline, postbaseline, and change from baseline in urine creatinine will be summarized by treatment group and visit using descriptive statistics. Baseline and change from baseline will be compared between the 2 treatment groups using a 2-sided Wilcoxon rank sum test.

## 7.2.5.3. Albuminuria by Quantitative Assessment

The baseline, postbaseline, changes from baseline, and percentage change from baseline in UACR will be summarized by treatment group and visit using descriptive statistics. Baseline and percentage change from baseline will be compared between the 2 treatment groups using a 2-sided Wilcoxon rank sum test.

The number and percentage of subjects with UACR  $< 30 \text{ mg/g versus} \ge 30 \text{ mg/g will be}$  summarized by baseline category at Weeks 24, 48, and based on the last on-treatment value (ie, data collected after the first dose date up to 1 day after the randomized phase last dose date) {KDIGO Guideline Development Staff 2013}.

Median (Q1, Q3) percentage change from baseline in UACR over time will be plotted by treatment group.

## 7.3. Body Weight, Height, and Vital Signs

Descriptive statistics will be provided by treatment group for vital signs and body weight as follows:

- Baseline values
- Values at each postbaseline analysis window
- Change from baseline at each postbaseline analysis window

A baseline value will be defined as the last nonmissing value obtained on or prior to the date of first dose of randomized study drug. Change from baseline to a postbaseline visit will be defined as the postbaseline value minus the baseline value.

In the case of multiple values in an analysis window, data will be selected for analysis as described in Section 3.8.3. No formal statistical testing is planned.

A by-subject listing of vital signs will be provided by subject ID number and visit in chronological order. In the same listing, a by-subject listing of body weight, height, and BMI will be provided.

## 7.4. Prior and Concomitant Medications

#### 7.4.1. Antiretroviral Medications

Any nonstudy ARV medications used prior to, during, or after the study (if collected) are all recorded on the ARV eCRF. All ARV medications recorded on the ARV eCRF will be coded using the Gilead-modified World Health Organization (WHO) Drug Dictionary for ARV medication. The WHO preferred name and drug code will be attached to the clinical database. All ARV medications recorded on the ARV eCRF will be listed. No inferential statistics will be provided.

#### 7.4.2. Prior Antiretroviral Medications

Prior ARV medications are defined as ARV medications taken on or up to 2 days prior to the first dose date of randomized study drug based on ARVs reported on ARV eCRF (see Appendix 5 for details). The number and percentage of subjects in each prior ARV regimen will be summarized as part of baseline disease characteristics table.

#### 7.4.3. Concomitant Non-Antiretroviral Medications

Concomitant non-ARV medications (ie, medications other than study drug that are taken while receiving study drug) will be coded using the WHO Drug Dictionary. The WHO preferred name and drug code will be attached to the clinical database. Use of concomitant medications from the randomized phase first dose date to the randomized phase last dose date will be summarized

(number and percentage of subjects) by treatment group and preferred name. Multiple drug use (by preferred name) will be counted only once per subject. The summary will be sorted by decreasing order of total frequency.

If the start or stop date of non-ARV medications is incomplete, the month and year (or year alone, if month is not recorded) of the start or stop date will be used to determine whether the non-ARVs are concomitant or not for the randomized phase of the study. The medication is concomitant if the month and year of the start or stop (or year of the start or stop, if month is not recorded) of the medication does not meet either of the following criteria:

- The month and year of start of the medication is after the randomized phase last dose date
- The month and year of stop of the medication is before the randomized phase first dose date

If the start and stop date of non-ARV medications are complete, the start date is not after the randomized phase last dose date and the stop date is not before the randomized phase first dose date, or the non-ARV medications are marked as ongoing and start date is on or before the randomized phase last dose date, the non-ARV medications are concomitant for the randomized phase of the study.

Summaries of non-ARV concomitant medications will be provided for the safety analysis set. Subjects with any non-ARV concomitant medications will be listed. No inferential statistics will be provided.

## 7.5. Electrocardiogram Results

A shift table of the investigators' assessment of ECG results at each scheduled postbaseline visit compared with baseline values will be presented by treatment group using the following categories: normal; abnormal, not clinically significant; abnormal, clinically significant; or missing. The number and percentage of subjects in each cross-classification group of the shift table will be presented. Subjects with a missing value at baseline or postbaseline will not be included in the denominator for percentage calculation. No inferential statistics will be provided.

A by-subject listing for ECG assessment results will be provided by subject ID number and visits in chronological order.

#### 7.6. Other Safety Measures

A data listing will be provided for subjects experiencing pregnancy during the study. Physical examination was not collected in the eCRF. Therefore, it will not be included in the analysis.

## 7.7. Subject Subgroup for Safety Endpoints

Incidence of all treatment-emergent AEs will be repeated within each subgroup defined in Section 3.4.2 using the safety analysis set. In addition, subgroup analysis by prior treatment regimen (ie, TDF-containing regimen versus non-TDF containing regimen) will be performed for renal endpoints including urine RBP to creatinine ratio, beta-2 microglobulin to creatinine ratio, and UACR

#### 7.8. Changes From Protocol-Specified Safety Analyses

No change from protocol-specified safety analysis is planned.

## 8. PHARMACOKINETIC ANALYSES

## 8.1. Analysis for Trough and Postdose PK (PK Analysis Set)

The following listings will be provided for trough and postdose PK analysis for subjects in the PK analysis set:

- Listing of PK sampling details ("Trough" PK samples [defined as samples collected within a range of 20.0 to 28.0 hours, inclusive, after previous dosing time] will be marked in the listing)
- Listing of study drug administration record for PK dosing

PK sampling details for single PK, trough PK, and postdose PK samples will be included in one listing. Similarly, study drug administration records for single PK, trough PK, and postdose PK samples will also be included in one listing.

## 8.2. Changes from Protocol-Specified Pharmacokinetic Analysis

No change from protocol-specified PK analyses is planned.

## 9. SPECIAL POPULATION ANALYSES

Only randomized phase data will be included for the special population analyses.

## 9.1. Analyses for HIV/HBV Coinfected Subjects

Subjects with HIV/HBV coinfection at baseline are defined as subjects meet any of the following two criteria:

- Positive HBsAg on or prior to the randomized phase first dose date, or
- Negative HBsAg, negative HBsAb, positive HBcAb, and quantifiable HBV DNA (ie, HBV DNA ≥ 20 IU/mL) on or prior to the randomized phase first dose date.

The following analyses will be provided by treatment and overall for subjects with HIV/HBV coinfection at baseline:

- The proportion of subjects with HBV DNA < 29 IU/mL at baseline and Week 48
- Treatment-emergent adverse events overall summary
- Treatment-emergent adverse events by SOC, HLT, and PT
- Treatment-emergent laboratory abnormalities
- The change from baseline for liver-related laboratory tests, including ALT, AST, ALP, total bilirubin, direct and indirect bilirubin
- Listing of adverse events
- Listing of liver-related laboratory tests and HBV DNA results

HBV DNA will be analyzed using observed, on-treatment data (ie, data collected up to the 1 day after the randomized phase last dose date) for subject in the FAS with HIV/HBV coinfection at baseline.

Subjects with incident HIV/HBV coinfection while on study drug (if any) are defined as subjects who are not HIV/HBV coinfected at baseline and meet any of the following criteria:

- Positive HBsAg after the randomized phase first dose date and on or prior to the randomized phase last dose date, or
- Negative HBsAg, negative HBsAb, positive HBcAb, and quantifiable HBV DNA (ie, HBV DNA ≥ 20 IU/mL) after the randomized phase first dose date and on or prior to the randomized phase last dose date, or

• Experience any of the following adverse events (ie, selected MedDRA PTs from the SMQ of "Liver Infections") after the randomized phase first dose date and on or prior to the randomized phase last dose date: Acute hepatitis B, Chronic hepatitis B, Congenital hepatitis B infection, Hepatitis B, Hepatitis B core antibody positive, Hepatitis B DNA assay positive, Hepatitis B surface antigen positive, Hepatitis B virus test positive.

The following listings will be provided for subjects with incident HIV/HBV coinfection while on study drug (if any):

- Listing of adverse events
- Listing of liver-related laboratory tests and HBV DNA results

## 9.2. Analyses for HIV/HCV Coinfected Subjects

Subjects with HIV/HCV coinfection at baseline are defined as subjects with positive HCV antibody (HCVAb) and quantifiable HCV RNA (ie, HCV RNA ≥ 15 IU/mL) on or prior to the randomized phase first dose date. The following analyses will be conducted for subjects with HIV/HCV coinfection at baseline:

- Treatment-emergent adverse events overall summary
- Treatment-emergent adverse events by SOC, HLT, and PT
- Treatment-emergent laboratory abnormalities
- Listing of adverse events
- Listing of liver-related laboratory tests and HCV RNA results

Subjects with incident HIV/HCV coinfection while on study drug are defined as subjects who are not HIV/HCV coinfected at baseline and meet any of the following criteria:

- Positive HCVAb after the randomized phase first dose date and on or prior to the randomized phase last dose date with baseline HCVAb Negative or missing, or
- Quantifiable HCV RNA (ie, HCV RNA ≥ 15 IU/mL) after the randomized phase first dose date and on or prior to the randomized phase last dose date, or
- Experience any of the following adverse events (ie, selected MedDRA PTs from the SMQ of "Liver Infections") after the randomized phase first dose date and on or prior to the randomized phase last dose date: Acute hepatitis C, Chronic hepatitis C, Hepatitis C, Hepatitis C antibody positive, Hepatitis C RNA positive, Hepatitis C virus test positive

The following listings will be provided for subjects with incident HIV/HCV coinfection while on study drug:

- Listing of adverse events
- Listing of liver-related laboratory tests and HCV RNA results

## 10. REFERENCES

- KDIGO Guideline Development Staff. KDIGO 2012 Clinical Practice Guideline for the Evaluation and Management of Chronic Kidney Disease. Kidney international. Supplement 2013;3 (1):v-150.
- U. S. Department of Health and Human Services, Food and Drug Administration (FDA), Center for Drug Evaluation and Research (CDER). Human Immunodeficiency Virus-1 Infection: Developing Antiretroviral Drugs for Treatment. Guidance for Industry. Silver Spring, MD. November, 2015.

## 11. SOFTWARE

SAS® Version 9.4 (SAS Institute Inc., Cary, NC, USA) is to be used for all programming of tables, listings, and figures.

nQuery Advisor® Version 6.0 (Statistical Solutions, Cork, Ireland) is to be used for sample size and power calculation.

Phoenix WinNonlin® Version 6.4 (Certara USA Inc., Princeton, NJ, USA) is to be used for all PK analyses.

# 12. SAP REVISION

| Revision Date<br>(dd month, yyyy) | Section | Summary of Revision | Reason for Revision |
|---|---|---|---|

#### 13. **APPENDICES**

| A | ppend | lix 1 | . S | tu | dy | Pr | oced | lures | Tab | le |
|---|-------|-------|-----|----|----|----|------|-------|-----|----|
|---|-------|-------|-----|----|----|----|------|-------|-----|----|

Appendix 1. Appendix 2. Appendix 3. Appendix 4. Appendix 5. Flowchart of US FDA-defined Snapshot Algorithm Selected Medical History

Hepatic Events

Programming Specification

**Appendix 1. Study Procedures Table** 

| | | | End of Week <sup>c</sup> | | Post Week 48 <sup>d,v</sup> | 30 Day | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| <b>Study Procedure</b> | Screeninga | Day 1 <sup>b</sup> | 4 | 8 | 12 | 24 | 36 | 48 | Every 12 Weeks | Follow-Up <sup>e</sup> | $ESDD^f$ |
| Informed Consent | X | | | | | | | | | | |
| Medical History | X | | | | | | | | | | |
| Concomitant Medications | X | X | X | X | X | X | X | X | X | X | X |
| Adverse Events | X | X | X | X | X | X | X | X | X | X | X |
| Complete Physical Exam | X | X | | | | X | | X | | | X |
| Symptom-Directed Physical Exam | | | X | X | X | | X | | X | X | |
| 12-Lead ECG | X | X | | | | X | | X | | | X |
| Height | X | | | | | | | | | | |
| Weight | X | X | X | X | X | X | X | X | X | X | X |
| Vital Signs <sup>g</sup> | X | X | X | X | X | X | X | X | X | X | X |
| Urinalysis | X | X | X | X | X | X | X | X | X | X | X |
| Urine Chemistry <sup>h</sup> | | X | | | | X | | X | X <sup>w</sup> | | |
| Urine Pregnancy Test <sup>i</sup> | | X | X | X | X | X | X | X | X | X | X |
| Serum Pregnancy Test <sup>i</sup> | X | | | | | | | | | | |
| Chemistry Profile <sup>j</sup> | X | X | X | X | X | X | X | X | X | X | X |
| Metabolic Assessments <sup>k</sup> | | X | | | X | X | | X | Xw | | |
| Estimated GFR | X | X | X | X | X | X | X | X | X | X | X |
| Hematology Profile <sup>1</sup> | X | X | X | X | X | X | X | X | X | X | X |
| Plasma HIV-1 RNA <sup>m</sup> | X | X | X | X | X | X | X | X | X | X | X |
| CD4+ Cell Count | X | X | X | X | X | X | X | X | X | X | X |
| HBV Blood Planel <sup>n</sup> | X | | | | | | | | | | |

| | | | End of Week <sup>c</sup> | | | | | | Post Week 48 <sup>d,v</sup> | 20 Day | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Procedure | Screening <sup>a</sup> | Day 1b | 4 | 8 | 12 | 24 | 36 | 48 | Every 12 Weeks | 30 Day<br>Follow-Up <sup>e</sup> | ESDD <sup>f</sup> |
| Plasma HBV DNA° | | X | | | X | X | | X | $X^{w}$ | Î | X |
| HCVAb <sup>p</sup> | X | 8 | | | | | | 8 8 | | | |
| HCV RNA <sup>p</sup> | X | \$ \$1 | | | 3 | X | | X | Xw | | |
| HIV-1 Genotype/Phenotype <sup>q</sup> | | | | | | | | $X^q$ | | | $X^q$ |
| Single PK Draw <sup>r</sup> | 2,0,3 | | | X | | X | X | 1d 6 | | | |
| Trough PK Draw <sup>s</sup> | | | X | | X | | | | | | |
| PK Sample (post-dose) <sup>s</sup> | | | X | | X | | | | | | |
| Observed In-Clinic Dose <sup>s</sup> | | | X | | X | | | | | | |
| Provide Dosing Diary <sup>u</sup> | | X | X | X | X | X | | | | | |
| Collect Dosing Diary <sup>x</sup> | | | X | X | X | X | X | | | | |
| Plasma Sample Storage <sup>t</sup> | | X | X | X | X | X | X | X | X | | X |
| Urine Sample Storage <sup>t</sup> | & p | X | X | X | X | X | X | X | X | | X |
| Whole Blood Storage Sample <sup>t</sup> | | X | | | | | | | | | |
| PPD | | X | | | | | | Lid b | | | |
| Randomization | | X | | | | | | | | | |
| Study Drug Dispensation | 7. C | X | X | X | X | X | X | $\mathbf{X}^{\mathbf{v}}$ | X <sup>v</sup> | | |
| Study Drug Accountability | | | X | X | X | X | X | X | X | | X |

a Evaluations to be completed within 30 days prior to Day 1.

b Subjects should initiate dosing of study drug on the same day as the Day 1 visit.

c All study visits should be ± 2 days of the protocol-specified visit date based on the Day 1 visit through Week 12 and completed within ± 6 days at Week 24 and Week 36, unless otherwise specified. The visit window at Week 48 will be ± 6 weeks of the protocol-specified visit date.

d At the Week 48 Visit, subjects in a country where GS-9883/F/TAF FDC is not available will be given the option to receive GS-9883/F/TAF FDC for an additional 48 weeks, or until the product becomes accessible to subjects through an access program, or until Gilead Sciences elects to discontinue the study in that country, whichever occurs first. Study visits are to be completed every 12 weeks, within ± 6 days of the protocol-specified visit date unless otherwise specified.

- e Must be completed 30 days after discontinuing study drug. For the purpose of scheduling a 30-Day Follow-Up Visit, a ± 6 days window may be used. Required for subjects who permanently discontinue study drug prior to Week 48 and do not continue in the study through at least one subsequent visit after the ESDD visit. Subjects who participate post Week 48 will be required to return to the clinic 30 days after the completion of study drugs for the 30-Day Follow-Up Visit.
- f Early Study Drug Discontinuation visit to occur within 72 hours of last dose of study drug. Subjects will be asked to continue attending the scheduled study visits through the Week 48 Visit even if the subject discontinues study drug.
- g Vital signs measurements including blood pressure, pulse, respiratory rate, and temperature
- h Urine Chemistry includes urine albumin, urine creatinine, urine protein, retinol binding protein, and beta-2 microglobulin
- i Women of childbearing potential only. Positive urine pregnancy tests will be confirmed with a serum test.
- j Chemistry profile: alkaline phosphatase, AST, ALT, GGT, total bilirubin, direct and indirect bilirubin, total protein, albumin, bicarbonate, BUN, calcium, chloride, creatinine, glucose, phosphorus, magnesium, potassium, sodium, uric acid, and amylase (reflex lipase testing is performed in subjects with total amylase > 1.5 × ULN). At Day 1, Weeks 24, and 48 and every 24 weeks during the post Week 48 period, analyses of glucose will be done as part of the fasting metabolic assessments and not as part of the chemistry profile. TSH will be collected at Screening, Day 1, Weeks 24, and 48, as well as every 24 weeks post Week 48, and ESDD if applicable.
- k Fasting glucose and lipid panel (total cholesterol, HDL, direct LDL, triglycerides). If the subject has not fasted prior to the visit, the visit may proceed, but the subject must return within 72 hours in a fasted state to draw blood for the metabolic assessments.
- 1 CBC with differential and platelet count.
- m If the HIV-1 RNA value is ≥ 50 copies/mL at Week 48, a retest HIV-1 RNA value must be collected within two to three weeks of the initial test.
- n Hepatitis B Virus (HBV) blood panel: Hepatitis B virus surface antigen (HBsAg), Hepatitis B virus surface antibody (HBsAb) and Hepatitis B virus core antibody (HBcAb). If positive HBsAg, reflex testing for plasma HBV DNA, HBeAg (if negative, reflex HBeAb), and quantitative HBsAg. If positive HBcAb with negative HBsAg and negative HBsAb, reflex testing for plasma HBV DNA (if positive, reflex HBeAg). If HBeAg is performed and found to be negative, reflex HBeAb.
- o For subjects who meet the definition of HBV infection, the following will be conducted by the central laboratory: HBsAb, HBsAg (qualitative and quantitative) and HBeAg (if negative, reflex HBeAb) at Days 1, 12, 24 and then every 24 weeks.
- p Subjects who are HCVAb positive will have a HCV RNA test performed at screening and every 24 weeks.
- q HIV-1 genotype/phenotype testing for subjects with HIV-1 RNA ≥ 200 copies/mL and virologic rebound, at early study drug discontinuation or Week 48. Following unconfirmed virologic rebound, subjects will be asked to return to the clinic (2-3 weeks later) prior to the next scheduled visit or at the next scheduled study visit, for a HIV-1 RNA and HIV-1 genotype/phenotype (reverse transcriptase, protease and integrase) blood draw. Based on the results of this testing, subjects should be managed according to the Virologic Rebound Schema (Section 6.13.1).
- r All subjects on GS-9883/F/TAF (Treatment Group 1 only) will have a single anytime PK blood sample collected at Weeks 8, 24 and 36.
- s Subjects on GS-9883/F/TAF (Treatment Group 1 only) will have a Trough PK blood sample collected between 20-28 hours following their last dose at Weeks 4 and 12. Subjects must be instructed to not take their study drugs on the morning of their visit for the trough sample collection. If the subject has taken their dose of study drugs prior to the visit, the visit may proceed, but the subject must return within 72 hours for the single trough PK blood sample collection. In the event a subject routinely takes their study drug in the evening, a single anytime sample may be drawn at Weeks 4 and 12 as the subject will not be instructed to change their dosing time to accommodate this trough PK draw. A post-dose PK blood sample will be collected between 1 and 4 hours post dose following an observed, in-clinic dose.
- t Plasma storage samples banked for possible future protocol-related testing (safety, virology, pharmacokinetic analysis). Urine storage samples banked for possible future protocol-related safety testing including urine chemistry. Whole blood sample for potential virologic resistance testing and/or HIV DNA genotyping.
- A dosing diary will be dispensed for all Treatment Group 1 subjects to complete prior to each of the PK sample visits.
- v Open-label GS-9883/F/TAF FDC will be dispensed to subjects participating in the study post Week 48 starting at the Week 48 Visit.
- w Every 24 weeks only.
- x Dosing diaries will be collected from subjects for the single anytime PK and trough PK collection (Treatment Group 1 only). If a dosing diary is not returned the site may ask the subject for the time of the last dose and if it was taken with or without food.

## Appendix 2. Flowchart of US FDA-defined Snapshot Algorithm

The following flowchart for US FDA-defined snapshot algorithm is based on the US FDA Guidance on Human Immunodeficiency Virus-1 Infection: Developing Antiretroviral Drugs for Treatment {U. S. Department of Health and Human Services 2015}



<sup>\*</sup> On-Treatment HIV-1 RNA data include all HIV-1 RNA data for subjects who are on-going and HIV-1 RNA data up to 1 day after the last dose date of study drug for subjects who prematurely discontinue or complete study drug.

## **Appendix 3. Selected Medical History**

Number and percentage of subjects with selected medical history of Diabetes Mellitus, Hypertension, Cardiovascular Disease, and Hyperlipidemia will be summarized by treatment as baseline disease characteristics. A subject who had medical history of one of these diseases is a subject who experience at least one of the following events:

- At least 1 medical history record with MedDRA PT (mh.MDRPT) in the following selected PT listing for the corresponding disease with start date on or prior to the randomized phase first dose date.
- At least 1 AE record with MedDRA PT (ae.MDRPT) in the following selected PT listing for the corresponding disease with start date on or prior to the randomized phase first dose date.
- At least 1 concomitant medications record with medication class and indication in the following selected listing for the corresponding disease with start date on or prior to the randomized phase first dose date.

If the start date is incomplete but the month and year (or year alone) of the start date is the same as or before the month and year (or year alone) of the first dosing date of randomized study drug, the event will be included. If the start date is completely missing, the event will be included.

Four variables (ie, DIABETES, HTENSION, CARDDIS, and HLIPDEM) will be added to raw Medical History and Adverse Events datasets. A medical history or an AE record will be flagged for a disease of interest if its MedDRA PT included in the following pre-specified PT list for the corresponding disease of interest, which include all PTs from the narrow or broad search of the following SMQs under MedDRA 19.1 provided by Gilead DSPH and reviewed by Gilead medical monitors.

| Disease of Interest | SMQ Source |
|---|---|
| Diabetes Mellitus (DIABETES) | Hyperglycaemia/new onset diabetes mellitus (SMQ) – Narrow Scope Term |
| Hyperlipidemia (HLIPDEM) | Dyslipidaemia (SMQ) |
| Hypertension (HTENSION) | Hypertension (SMQ) |
| Cardiovascular disease (CARDDIS) | Ischaemic central nervous system vascular conditions (SMQ) – Narrow Scope Term |
| | Myocardial infarction (SMQ) - Narrow Scope Term |
| | Other ischaemic heart disease (SMQ) - Narrow Scope Term |

Similarly, two variables (ie, DRUGF and DRUGTYP) will be added to raw Concomitant Medication dataset. A concomitant medication record will be flagged for a disease of interest if its medication class and indication included in the following listing for the corresponding disease of interest.

The selected combination of medication class and indication are listed as follows, which was reviewed by Gilead medical monitors.

| | <b>Medication Class (WHOATC2)</b> | Indication (CMINDC) | WHOGEN |
|---|---|---|---|
| Нур | ertension (HTENSION) | | |
| 1 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | | LISINOPRIL |
| 2 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ANTI-HYPERTENSIVE | LOSARTAN |
| 3 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ARTERIAL HYPENTENSION | RAMIPRIL |
| 4 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ARTERIAL HYPERTENSION | CAPTOPRIL |
| 5 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ARTERIAL HYPERTENSION | ENALAPRIL |
| 6 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ARTERIAL HYPERTENSION | HYDROCHLOROTHIAZIDE<br>W/OLMESARTAN |
| 7 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ARTERIAL HYPERTENSION | OLMESARTAN MEDOXOMIL |
| 8 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ARTERIAL HYPERTENSION | RAMIPRIL |
| 9 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ARTERIAL HYPERTENSION | SALUTEC |
| 10 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ARTERIAL HYPERTENSION | VALSARTAN |
| 11 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ARTERIAL HYPERTENSION<br>STAGE I | CAPTOPRIL |
| 12 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ARTERIAL HYPERTENSION<br>STAGE 1 | CANDESARTAN |
| 13 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | BENIGN ESSENTIAL<br>HYPERTENSION | LISINOPRIL |
| 14 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | BENIGN ESSENTIAL<br>HYPERTENSION | LOSARTAN |
| 15 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ESSENTIAL<br>(PRIMARY)HYPERTESION | ZESTORETIC |
| 16 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ESSENTIAL HYPERTENSION | COROVAL B |
| 17 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ESSENTIAL HYPERTENSION | ENALAPRIL MALEATE |
| 18 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ESSENTIAL HYPERTENSION | LISINOPRIL |
| 19 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ESSENTIAL HYPERTENSION | LOSARTAN |
| 20 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ESSENTIAL HYPERTENSION | TRIBENZOR |
| 21 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ESSENTIAL HYPERTENSION | ZESTORETIC |
| 22 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ESSENTIAL PRIMARY<br>HYPERTENSION | IRBESARTAN |
| 23 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HIGH BLOOD PRESSURE | COVERAM |

| | Medication Class (WHOATC2) | Indication (CMINDC) | WHOGEN |
|---|---|---|---|
| 24 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HIGH BLOOD PRESSURE | ENALAPRIL |
| 25 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HIGH BLOOD PRESSURE | IRBESARTAN |
| 26 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HIGH BLOOD PRESSURE | LISINOPRIL |
| 27 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HIGH BLOOD PRESSURE | LOSARTAN |
| 28 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HIGH BLOOD PRESSURE | LOSARTAN POTASSIUM |
| 29 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HIGH BLOOD PRESSURE | RAMIPRIL |
| 30 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HIGH BOLD PRESSURE | LOSARTAN |
| 31 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HISTORY OF MYOCARDITIS | RAMIPRIL |
| 32 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HTN | ZESTORETIC |
| 33 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERRTENSION | ZESTORETIC |
| 34 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTEENSION | LISINOPRIL |
| 35 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | AMLODIPINE<br>W/HYDROCHLOROTHIAZIDE/VALS<br>ARTAN |
| 36 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | AMLODIPINE W/VALSARTAN |
| 37 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | BENAZEPRIL |
| 38 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | BENAZEPRIL HYDROCHLORIDE |
| 39 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | BENICAR HCT |
| 40 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | BI PREDONIUM |
| 41 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | CANDESARTAN |
| 42 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | CANDESARTAN CILEXETIL |
| 43 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | CAPTOPRIL |
| 44 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | CO-DIOVAN |
| 45 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | COROVAL B |
| 46 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | DIOVAN AMLO |

| | Medication Class (WHOATC2) | Indication (CMINDC) | WHOGEN |
|---|---|---|---|
| 47 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | DIOVAN TRIPLE |
| 48 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | EDARBYCLOR |
| 49 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | ENALAPRIL |
| 50 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | ENALAPRIL MALEATE |
| 51 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | FOSINOPRIL |
| 52 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | HYDROCHLOROTHIAZIDE<br>W/LOSARTAN |
| 53 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | HYZAAR |
| 54 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | IRBESARTAN |
| 55 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | KARVEA HCT |
| 56 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | LISINOPRIL |
| 57 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | LOSARTAN |
| 58 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | LOSARTAN POTASSIUM |
| 59 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | NAPRIX A |
| 60 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | OLMESARTAN MEDOXOMIL |
| 61 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | PERINDOPRIL ERBUMINE |
| 62 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | PRITORPLUS |
| 63 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | QUINAPRIL |
| 64 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | RAMIPRIL |
| 65 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | SALUTEC |
| 66 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | TELMISARTAN |
| 67 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | TRIBENZOR |
| 68 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | VALSARTAN |
| 69 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | VASERETIC |
| 70 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION | ZESTORETIC |

| | Medication Class (WHOATC2) | Indication (CMINDC) | WHOGEN |
|---|---|---|---|
| 71 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION ESSENTIAL | CANDESARTAN CILEXETIL |
| 72 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION ESSENTIAL | DIOVAN TRIPLE |
| 73 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION, BENIGN | LISINOPRIL |
| 74 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION, BILATERAL<br>LOWER LEG SWELLING | LISINOPRIL |
| 75 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION, ESSENTIAL | ZESTORETIC |
| 76 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION, WORSENING HYPERTENSION | LISINOPRIL |
| 77 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSIONPROPHYLAXI<br>S | RAMIPRIL |
| 78 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSIVE | RAMIPRIL |
| 79 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSIVE CRISIS | CAPTOPRIL |
| 80 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENTION | LISINOPRIL |
| 81 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTONIA | RAMIPRIL |
| 82 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPOKALEMIA | LOSARTAN POTASSIUM |
| 83 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | POOR CONTROL OF BLOOD<br>PRESSURE | LISINOPRIL |
| 84 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | PREVENTATIVE FOLLOWING<br>ACUTE MYCARDIAL<br>INFARCTION | PERINDOPRIL |
| 85 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | PRIMARY ESSENTIAL<br>HYPERTENSION | ENALAPRIL MALEATE |
| 86 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | PROTEINURIA | BENAZEPRIL |
| 87 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | PROTEINURIA | ENALAPRIL |
| 88 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | PROTEINURIA | LISINOPRIL |
| 89 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | WORSENING HYPERTENSION | BENAZEPRIL |
| 90 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | WORSENING HYPERTENSION | PERINDOPRIL |
| 91 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | WORSENING HYPERTENSION | PRETERAX ARGININE |
| 92 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | WORSENING OF<br>HYPERTENSION | LISINOPRIL |
| 93 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | WORSENING OF<br>HYPERTENSION | RAMIPRIL |

| | Medication Class (WHOATC2) | Indication (CMINDC) | WHOGEN |
|---|---|---|---|
| 94 | ANTIHYPERTENSIVES | BENIGN HIGH BLOOD<br>PRESSURE | DOXAZOSIN |
| | AWITHTERTERSIVES | EXACERBATION OF | DOMEOSIN |
| 95 | ANTIHYPERTENSIVES | HYPERTENSION | CLONIDINE |
| 96 | ANTIHYPERTENSIVES | HEADACHE | HYDRALAZINE |
| 97 | ANTIHYPERTENSIVES | HIGH BLOOD PRESSURE | CLONIDINE HYDROCHLORIDE |
| 98 | ANTIHYPERTENSIVES | HIGH BLOOD PRESSURE | RILMENIDINE |
| 99 | ANTIHYPERTENSIVES | HYPERTENSION | CLONIDINE |
| 100 | ANTIHYPERTENSIVES | HYPERTENSION | CLONIDINE HYDROCHLORIDE |
| 101 | ANTIHYPERTENSIVES | HYPERTENSION | DOXAZOSIN |
| 102 | ANTIHYPERTENSIVES | HYPERTENSION | DOXAZOSIN MESILATE |
| 103 | ANTIHYPERTENSIVES | HYPERTENSION | HYDRALAZINE |
| 104 | ANTIHYPERTENSIVES | HYPERTENSION | HYDRALAZINE HYDROCHLORIDE |
| 105 | ANTIHYPERTENSIVES | HYPERTENSION | METHYLDOPA |
| 106 | ANTIHYPERTENSIVES | HYPERTENSION | TADALAFIL |
| 107 | ANTIHYPERTENSIVES | PULMONARY HYPERTENSION | TADALAFIL |
| 108 | ANTIHYPERTENSIVES | VASODILATION-STENT<br>PROCEDURE | HYDRALAZINE |
| 109 | ANTIHYPERTENSIVES | WORSENING HYPERTENSION | HYDRALAZINE HYDROCHLORIDE |
| 110 | BETA BLOCKING AGENTS | ARTERIAL HYPERTENSION | ATENOLOL |
| 111 | BETA BLOCKING AGENTS | ARTERIAL HYPERTENSION | METOPROLOL SUCCINATE |
| 112 | BETA BLOCKING AGENTS | ARTERIAL HYPERTENSION / ICHEMIC HEART DISEASE | BISOPROLOL |
| 113 | BETA BLOCKING AGENTS | ESSENTIAL HYPERTENSION | METOPROLOL |
| 114 | BETA BLOCKING AGENTS | HEART FAILURE AND<br>HYPERTENSION | CARVEDILOL |
| 115 | BETA BLOCKING AGENTS | HEART HEALTH | ATENOLOL |
| 116 | BETA BLOCKING AGENTS | HIGH BLOOD PRESSURE | ATENOLOL |
| 117 | BETA BLOCKING AGENTS | HIGH BLOOD PRESSURE | BISOPROLOL<br>W/HYDROCHLOROTHIAZIDE |
| 118 | BETA BLOCKING AGENTS | HIGH BLOOD PRESSURE | METOPROLOL |
| 119 | BETA BLOCKING AGENTS | HISTORY OF MYOCARDITIS | BISOPROLOL |
| 120 | BETA BLOCKING AGENTS | HYPERTENSION | ATENOLOL |
| 121 | BETA BLOCKING AGENTS | HYPERTENSION | BISOPROLOL FUMARATE |
| 122 | BETA BLOCKING AGENTS | HYPERTENSION | CARVEDILOL |
| 123 | BETA BLOCKING AGENTS | HYPERTENSION | LABETALOL |
| 124 | BETA BLOCKING AGENTS | HYPERTENSION | METOPROLOL |
| 125 | BETA BLOCKING AGENTS | HYPERTENSION | METOPROLOL SUCCINATE |
| 126 | BETA BLOCKING AGENTS | HYPERTENSION | METOPROLOL TARTRATE |
| 127 | BETA BLOCKING AGENTS | HYPERTENSION | NEBICARD V |
| 128 | BETA BLOCKING AGENTS | HYPERTENSION | NEBICARD-H |
| 129 | BETA BLOCKING AGENTS | HYPERTENSION | NEBIVOLOL |
| 130 | BETA BLOCKING AGENTS | HYPERTENSION | NEBIVOLOL HYDROCHLORIDE |

| | Medication Class (WHOATC2) | Indication (CMINDC) | WHOGEN |
|---|---|---|---|
| 131 | BETA BLOCKING AGENTS | HYPERTENSION | PROPRANOLOL |
| 132 | BETA BLOCKING AGENTS | HYPERTENSION | PROPRANOLOL HYDROCHLORIDE |
| 133 | BETA BLOCKING AGENTS | HYPERTENSION AND<br>MIGRAINE | ATENOLOL |
| 134 | BETA BLOCKING AGENTS | HYPERTENSION ESSENTIAL | ATENOLOL |
| 135 | BETA BLOCKING AGENTS | HYPERTENTION | METOPROLOL SUCCINATE |
| 136 | BETA BLOCKING AGENTS | HYPETENSION | BISOPROLOL |
| 137 | BETA BLOCKING AGENTS | PAROXYSM OF SINUS<br>TACHYCARDIA | PROPRANOLOL |
| 138 | BETA BLOCKING AGENTS | PRIMARY ESSENTIAL<br>HYPERTENSION | CARVEDILOL |
| 139 | BETA BLOCKING AGENTS | RAPID HEART BEAT | METOPROLOL SUCCINATE |
| 140 | CALCIUM CHANNEL BLOCKERS | ANTIHYPERTENSIVE | AMLODIPINE |
| 141 | CALCIUM CHANNEL BLOCKERS | ARTERIAL HYPERTENSION | AMLODIPINE |
| 142 | CALCIUM CHANNEL BLOCKERS | ARTERIAL HYPERTENSION | VERAPAMIL |
| 143 | CALCIUM CHANNEL BLOCKERS | ATRIAL FIBRILLATION | DILTIAZEM |
| 144 | CALCIUM CHANNEL BLOCKERS | ELEVATED BLOOD PRESSURE | AMLODIPINE |
| 145 | CALCIUM CHANNEL BLOCKERS | ELEVATED BLOOD PRESSURE | AMLODIPINE BESILATE |
| 146 | CALCIUM CHANNEL BLOCKERS | ESSENTIAL HYPERTENSION | AMLODIPINE |
| 147 | CALCIUM CHANNEL BLOCKERS | ESSENTIAL HYPERTENSION | AMLODIPINE BESILATE |
| 148 | CALCIUM CHANNEL BLOCKERS | ESSENTIAL HYPERTENSION | FELODIPINE |
| 149 | CALCIUM CHANNEL BLOCKERS | ESSENTIAL PRIMARY<br>HYPERTENSION | AMLODIPINE |
| 150 | CALCIUM CHANNEL BLOCKERS | HIGH BLOOD PRESSURE | AMLODIPINE |
| 151 | CALCIUM CHANNEL BLOCKERS | HTN | AMLODIPINE |
| 152 | CALCIUM CHANNEL BLOCKERS | HYPERTENSION | AMLODIPINE |
| 153 | CALCIUM CHANNEL BLOCKERS | HYPERTENSION | AMLODIPINE BESILATE |
| 154 | CALCIUM CHANNEL BLOCKERS | HYPERTENSION | BARNIDIPINE HYDROCHLORIDE |
| 155 | CALCIUM CHANNEL BLOCKERS | HYPERTENSION | DILTIAZEM |
| 156 | CALCIUM CHANNEL BLOCKERS | HYPERTENSION | DILTIAZEM HYDROCHLORIDE |
| 157 | CALCIUM CHANNEL BLOCKERS | HYPERTENSION | FELODIPINE |
| 158 | CALCIUM CHANNEL BLOCKERS | HYPERTENSION | NIFEDIPINE |
| 159 | CALCIUM CHANNEL BLOCKERS | HYPERTENSION | VERAPAMIL |
| 160 | CALCIUM CHANNEL BLOCKERS | HYPERTENSION<br>(ESSENTIAL/PRIMARY) | VERAPAMIL HYDROCHLORIDE |
| 161 | CALCIUM CHANNEL BLOCKERS | HYPERTENSION ESSENTIAL | FELODIPINE |
| 162 | CALCIUM CHANNEL BLOCKERS | HYPERTNESION | AMLODIPINE BESILATE |
| 163 | CALCIUM CHANNEL BLOCKERS | HYPTERTENSION | AMLODIPINE |
| 164 | CALCIUM CHANNEL BLOCKERS | PRESTUDY HYPERTENSION | AMLODIPINE |
| 165 | CALCIUM CHANNEL BLOCKERS | SECONDARY STROKE<br>PREVENTION | AMLODIPINE |
| 166 | CALCIUM CHANNEL BLOCKERS | SICK SINUS SYNDROME | VERAPAMIL |

| | Medication Class (WHOATC2) | Indication (CMINDC) | WHOGEN |
|---|---|---|---|
| | | WORSENING OF | |
| 167 | CALCIUM CHANNEL BLOCKERS | HYPERTENSION | AMLODIPINE |
| 168 | CARDIAC THERAPY | HYPERTENSION | UBIDECARENONE |
| 169 | DIURETICS | ARTERIAL HYPERTENSION | HYDROCHLOROTHIAZIDE |
| 170 | DIURETICS | BENIGN ESSENTIAL<br>HYPERTENSION | HYDROCHLOROTHIAZIDE |
| 171 | DIURETICS | BORDERLINE HYPERTENSION | HYDROCHLOROTHIAZIDE |
| 172 | DIURETICS | DIURETIC | FUROSEMIDE |
| 172 | DHIDETICS | ELEVATED BLOOD-PRESSURE<br>READING, WITHOUT<br>DIAGNOSIS OF | HWDDOCHI ODOTHIA ZIDE |
| 173 | DIURETICS | HYPERTENSION | HYDROCHLOROTHIAZIDE |
| 174 | DIURETICS | ESSENTIAL HYPERTENSION | FUROSEMIDE |
| 175 | DIURETICS | ESSENTIAL HYPERTENSION | HYDROCHLOROTHIAZIDE |
| 176 | DIURETICS | HIGH BLOOD PRESSURE | HYDROCHLOROTHIAZIDE |
| 177 | DIURETICS | HYPERTENSION | AMILORIDE |
| 178 | DIURETICS | HYPERTENSION | BUMETANIDE |
| 179 | DIURETICS | HYPERTENSION | CHLORTALIDONE |
| 180 | DIURETICS | HYPERTENSION | DYAZIDE |
| 181 | DIURETICS | HYPERTENSION | FUROSEMIDE |
| 182 | DIURETICS | HYPERTENSION | HYDROCHLOROTHIAZIDE |
| 183 | DIURETICS | HYPERTENSION | INDAPAMIDE |
| 184 | DIURETICS | HYPERTENSION | MODURETIC |
| 185 | DIURETICS | HYPERTENSION | SPIRONOLACTONE |
| 186 | DIURETICS | HYPERTENSION | TRIAMTERENE |
| 187 | DIURETICS | HYPERTENSION, BENIGN | HYDROCHLOROTHIAZIDE |
| 188 | DIURETICS | HYPERTENTION | HYDROCHLOROTHIAZIDE |
| 189 | DIURETICS | WORSENING HYPERTENSION | HYDROCHLOROTHIAZIDE |
| 190 | LIPID MODIFYING AGENTS | HIGH BLOOD PRESSURE | PRAVASTATIN |
| 191 | LIPID MODIFYING AGENTS | HIGH BLOOD PRESSURE | PRAVASTATIN SODIUM |
| Diab | etes Mellitus (DIABETES) | | |
| 1 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | DIABETES MELLITUS TYPE II | LISINOPRIL |
| 2 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | TYPE 2 DIABETES | LISINOPRIL |
| 3 | ANTIHYPERTENSIVES | UNCONTROLLED DIABETES<br>MELLITUS 2 | CLONIDINE HYDROCHLORIDE |
| 4 | ANTIHYPERTENSIVES | UNCONTROLLED DIABETES MELLITUS 2 | HYDRALAZINE HYDROCHLORIDE |
| 5 | BETA BLOCKING AGENTS | TYPE 2 DIABETES | METOPROLOL TARTRATE |
| 6 | DRUGS USED IN DIABETES | BORDERLINE DIABETES | METFORMIN |
| 7 | DRUGS USED IN DIABETES | DIABETES | DULAGLUTIDE |
| 8 | DRUGS USED IN DIABETES | DIABETES | GLIBENCLAMIDE |

| | Medication Class (WHOATC2) | Indication (CMINDC) | WHOGEN |
|---|---|---|---|
| 9 | DRUGS USED IN DIABETES | DIABETES | GLICLAZIDE |
| 10 | DRUGS USED IN DIABETES | DIABETES | GLIMEPIRIDE |
| 11 | DRUGS USED IN DIABETES | DIABETES | GLIPIZIDE |
| 12 | DRUGS USED IN DIABETES | DIABETES | HUMAN MIXTARD |
| 13 | DRUGS USED IN DIABETES | DIABETES | INSULIN |
| 14 | DRUGS USED IN DIABETES | DIABETES | INSULIN ASPART |
| 15 | DRUGS USED IN DIABETES | DIABETES | INSULIN DETEMIR |
| 16 | DRUGS USED IN DIABETES | DIABETES | INSULIN GLARGINE |
| 17 | DRUGS USED IN DIABETES | DIABETES | INSULIN HUMAN |
| 18 | DRUGS USED IN DIABETES | DIABETES | INSULIN LISPRO |
| 19 | DRUGS USED IN DIABETES | DIABETES | METAGLIP |
| 20 | DRUGS USED IN DIABETES | DIABETES | METFORMIN |
| 21 | DRUGS USED IN DIABETES | DIABETES | METFORMIN HYDROCHLORIDE |
| 22 | DRUGS USED IN DIABETES | DIABETES | PIOGLITAZONE |
| 23 | DRUGS USED IN DIABETES | DIABETES | PIOGLITAZONE HYDROCHLORIDE |
| 24 | DRUGS USED IN DIABETES | DIABETES | SITAGLIPTIN |
| 25 | DRUGS USED IN DIABETES | DIABETES - TYPE I | INSULIN GLARGINE |
| 26 | DRUGS USED IN DIABETES | DIABETES - TYPE I | INSULIN LISPRO |
| 27 | DRUGS USED IN DIABETES | DIABETES 2 | GLICLAZIDE |
| 28 | DRUGS USED IN DIABETES | DIABETES II | METFORMIN |
| 29 | DRUGS USED IN DIABETES | DIABETES KETOACIDOSIS | INSULIN |
| 30 | DRUGS USED IN DIABETES | DIABETES MELL. TYPE 2 | INSULIN DETEMIR |
| 31 | DRUGS USED IN DIABETES | DIABETES MELL. TYPE 2 | INSULIN LISPRO |
| 32 | DRUGS USED IN DIABETES | DIABETES MELL. TYPE 2 | METFORMIN |
| 33 | DRUGS USED IN DIABETES | DIABETES MELLITIS TYPE 2 | EMPAGLIFLOZIN |
| 34 | DRUGS USED IN DIABETES | DIABETES MELLITIS TYPE 2 | GLIBENCLAMIDE |
| 35 | DRUGS USED IN DIABETES | DIABETES MELLITIS TYPE 2 | INSULIN DETEMIR |
| 36 | DRUGS USED IN DIABETES | DIABETES MELLITIS TYPE 2 | INSULIN LISPRO |
| 37 | DRUGS USED IN DIABETES | DIABETES MELLITUS | DULAGLUTIDE |
| 38 | DRUGS USED IN DIABETES | DIABETES MELLITUS | EXENATIDE |
| 39 | DRUGS USED IN DIABETES | DIABETES MELLITUS | GLIPIZIDE |
| 40 | DRUGS USED IN DIABETES | DIABETES MELLITUS | HUMAN MIXTARD |
| 41 | DRUGS USED IN DIABETES | DIABETES MELLITUS | INSULIN ASPART |
| 42 | DRUGS USED IN DIABETES | DIABETES MELLITUS | INSULIN DETEMIR |
| 43 | DRUGS USED IN DIABETES | DIABETES MELLITUS | INSULIN GLARGINE |
| 44 | DRUGS USED IN DIABETES | DIABETES MELLITUS | INSULIN HUMAN |
| 45 | DRUGS USED IN DIABETES | DIABETES MELLITUS | INSULIN LISPRO |
| 46 | DRUGS USED IN DIABETES | DIABETES MELLITUS | LIRAGLUTIDE |
| 47 | DRUGS USED IN DIABETES | DIABETES MELLITUS | METFORMIN |
| 48 | DRUGS USED IN DIABETES | DIABETES MELLITUS | METFORMIN HYDROCHLORIDE |
| 49 | DRUGS USED IN DIABETES | DIABETES MELLITUS | RISTFOR |

| | Medication Class (WHOATC2) | Indication (CMINDC) | WHOGEN |
|---|---|---|---|
| 50 | DRUGS USED IN DIABETES | DIABETES MELLITUS | SITAGLIPTIN PHOSPHATE |
| 51 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYP II | INSULIN LISPRO |
| 52 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYP II | VELMETIA |
| 53 | DRUGS USED IN DIABETES | DIABETES MELLITUS 1 | INSULIN GLARGINE |
| 54 | DRUGS USED IN DIABETES | DIABETES MELLITUS 1 | INSULIN LISPRO |
| 55 | DRUGS USED IN DIABETES | DIABETES MELLITUS 11 | GLIPIZIDE |
| 56 | DRUGS USED IN DIABETES | DIABETES MELLITUS 2 | CANAGLIFLOZIN |
| 57 | DRUGS USED IN DIABETES | DIABETES MELLITUS 2 | DULAGLUTIDE |
| 58 | DRUGS USED IN DIABETES | DIABETES MELLITUS 2 | EXENATIDE |
| 59 | DRUGS USED IN DIABETES | DIABETES MELLITUS 2 | GLIBOMET |
| 60 | DRUGS USED IN DIABETES | DIABETES MELLITUS 2 | GLIMEPIRIDE |
| 61 | DRUGS USED IN DIABETES | DIABETES MELLITUS 2 | GLIPIZIDE |
| 62 | DRUGS USED IN DIABETES | DIABETES MELLITUS 2 | HUMAN MIXTARD |
| 63 | DRUGS USED IN DIABETES | DIABETES MELLITUS 2 | INSULIN ASPART |
| 64 | DRUGS USED IN DIABETES | DIABETES MELLITUS 2 | INSULIN DETEMIR |
| 65 | DRUGS USED IN DIABETES | DIABETES MELLITUS 2 | INSULIN GLARGINE |
| 66 | DRUGS USED IN DIABETES | DIABETES MELLITUS 2 | METFORMIN |
| 67 | DRUGS USED IN DIABETES | DIABETES MELLITUS 2 | METFORMIN HYDROCHLORIDE |
| 68 | DRUGS USED IN DIABETES | DIABETES MELLITUS II | GLIPIZIDE |
| 69 | DRUGS USED IN DIABETES | DIABETES MELLITUS II | METFORMIN |
| 70 | DRUGS USED IN DIABETES | DIABETES MELLITUS II | SITAGLIPTIN |
| 71 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYP 2 | METFORMIN |
| 72 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE 2 | GLIPIZIDE |
| 73 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE 2 | INSULIN GLARGINE |
| 74 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE 2 | INSULIN LISPRO |
| 75 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE 2 | METFORMIN |
| 76 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE 2 | METFORMIN HYDROCHLORIDE |
| 77 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE 2 | SITAGLIPTIN PHOSPHATE |
| 78 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE II | CANAGLIFLOZIN W/METFORMIN<br>HYDROCHLORIDE |
| 79 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE II | DULAGLUTIDE |
| 80 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE II | GLIPIZIDE |
| 81 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE II | HUMAN MIXTARD |
| 82 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE II | INSULIN |
| 83 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE II | INSULIN ASPART |
| 84 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE II | INSULIN DETEMIR |
| 85 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE II | INSULIN GLARGINE |
| 86 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE II | INSULIN LISPRO |
| 87 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE II | METFORMIN |
| 88 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE II | METFORMIN HYDROCHLORIDE |
| 89 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE II | NATEGLINIDE |

| | Medication Class (WHOATC2) | Indication (CMINDC) | WHOGEN |
|---|---|---|---|
| 90 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE II | SITAGLIPTIN PHOSPHATE |
| 91 | DRUGS USED IN DIABETES | DIABETES MELLITUS, TYPE II | METFORMIN HYDROCHLORIDE |
| 92 | DRUGS USED IN DIABETES | DIABETES TYPE 2 | GLIPIZIDE |
| 93 | DRUGS USED IN DIABETES | DIABETES TYPE 2 | HUMAN MIXTARD |
| 94 | DRUGS USED IN DIABETES | DIABETES TYPE 2 | INSULIN ASPART |
| 95 | DRUGS USED IN DIABETES | DIABETES TYPE 2 | INSULIN DETEMIR |
| 96 | DRUGS USED IN DIABETES | DIABETES TYPE 2 | INSULIN GLARGINE |
| 97 | DRUGS USED IN DIABETES | DIABETES TYPE 2 | INSULIN LISPRO |
| 98 | DRUGS USED IN DIABETES | DIABETES TYPE 2 | KOMBIGLYZE |
| 99 | DRUGS USED IN DIABETES | DIABETES TYPE 2 | METFORMIN |
| 100 | DRUGS USED IN DIABETES | DIABETES TYPE 2 | SITAGLIPTIN PHOSPHATE |
| 101 | DRUGS USED IN DIABETES | DIABETES TYPE II | METFORMIN |
| 102 | DRUGS USED IN DIABETES | DIABETES, TYPE 2 | GLIMEPIRIDE |
| 103 | DRUGS USED IN DIABETES | DIABETES, TYPE 2 | LIRAGLUTIDE |
| 104 | DRUGS USED IN DIABETES | DIABETES, TYPE 2 | PIOGLITAZONE |
| 105 | DRUGS USED IN DIABETES | DIABETIS | INSULIN GLARGINE |
| 106 | DRUGS USED IN DIABETES | DM2 | GLIPIZIDE |
| 107 | DRUGS USED IN DIABETES | DM2 | METFORMIN HYDROCHLORIDE |
| 108 | DRUGS USED IN DIABETES | HYPERGLICEMIA | GLIPIZIDE |
| 109 | DRUGS USED IN DIABETES | HYPERGLYCEMIA | INSULIN HUMAN |
| 110 | DRUGS USED IN DIABETES | HYPERGLYCEMIA | METFORMIN |
| 111 | DRUGS USED IN DIABETES | HYPERGLYCEMIA | METFORMIN HYDROCHLORIDE |
| 112 | DRUGS USED IN DIABETES | HYPERINSULINISM | METFORMIN |
| 113 | DRUGS USED IN DIABETES | HYPERTENSION | METFORMIN |
| 114 | DRUGS USED IN DIABETES | NONALCOHOLIC<br>STEATOHEPATITIS | METFORMIN |
| 115 | DRUGS USED IN DIABETES | TYPE 1 DIABETES | INSULIN DEGLUDEC |
| 116 | DRUGS USED IN DIABETES | TYPE 1 DIABETES MELLITUS | INSULIN ASPART |
| 117 | DRUGS USED IN DIABETES | TYPE 1 DIABETES MELLITUS | INSULIN GLARGINE |
| 118 | DRUGS USED IN DIABETES | TYPE 2 DIABETES | GLICLAZIDE |
| 119 | DRUGS USED IN DIABETES | TYPE 2 DIABETES | HUMAN MIXTARD |
| 120 | DRUGS USED IN DIABETES | TYPE 2 DIABETES | INSULIN ASPART |
| 121 | DRUGS USED IN DIABETES | TYPE 2 DIABETES | INSULIN GLARGINE |
| 122 | DRUGS USED IN DIABETES | TYPE 2 DIABETES | INSULIN LISPRO |
| 123 | DRUGS USED IN DIABETES | TYPE 2 DIABETES | METFORMIN |
| 124 | DRUGS USED IN DIABETES | TYPE 2 DIABETES | METFORMIN HYDROCHLORIDE |
| 125 | DRUGS USED IN DIABETES | TYPE 2 DIABETES | SITAGLIPTIN PHOSPHATE |
| 126 | DRUGS USED IN DIABETES | TYPE 2 DIABETES MELLITUS | GLIMEPIRIDE |
| 127 | DRUGS USED IN DIABETES | TYPE 2 DIABETES MELLITUS | HUMAN MIXTARD |
| 128 | DRUGS USED IN DIABETES | TYPE 2 DIABETES MELLITUS | INSULIN HUMAN |
| 129 | DRUGS USED IN DIABETES | TYPE 2 DIABETES MELLITUS | LIRAGLUTIDE |

| | Medication Class (WHOATC2) | Indication (CMINDC) | WHOGEN |
|---|---|---|---|
| 130 | DRUGS USED IN DIABETES | TYPE 2 DIABETES MELLITUS | METFORMIN HYDROCHLORIDE |
| 131 | DRUGS USED IN DIABETES | TYPE 2 DIABETES MELLITUS | PIOGLITAZONE |
| 132 | DRUGS USED IN DIABETES | TYPE II DIABETES | CANAGLIFLOZIN W/METFORMIN<br>HYDROCHLORIDE |
| 133 | DRUGS USED IN DIABETES | TYPE II DIABETES | DAPAGLIFLOZIN PROPANEDIOL<br>MONOHYDRATE W/METFO |
| 134 | DRUGS USED IN DIABETES | TYPE II DIABETES | GLIPIZIDE |
| 135 | DRUGS USED IN DIABETES | TYPE II DIABETES | INSULIN |
| 136 | DRUGS USED IN DIABETES | TYPE II DIABETES | INSULIN DETEMIR |
| 137 | DRUGS USED IN DIABETES | TYPE II DIABETES | INSULIN GLARGINE |
| 138 | DRUGS USED IN DIABETES | TYPE II DIABETES | LIRAGLUTIDE |
| 139 | DRUGS USED IN DIABETES | TYPE II DIABETES | METFORMIN |
| 140 | DRUGS USED IN DIABETES | TYPE II DIABETES | SITAGLIPTIN PHOSPHATE |
| 141 | DRUGS USED IN DIABETES | TYPE II DIABETES MELLITUS | EXENATIDE |
| 142 | DRUGS USED IN DIABETES | TYPE II DIABETES MELLITUS | METFORMIN |
| 143 | DRUGS USED IN DIABETES | TYPE II DIABETES MELLITUS | METFORMIN HYDROCHLORIDE |
| 144 | DRUGS USED IN DIABETES | UNCONTROLLED DIABETES MELLITUS 2 | INSULIN LISPRO |
| 145 | DRUGS USED IN DIABETES | UNCONTROLLED DIABETES<br>MELLITUS WITH<br>HYPERGLICEMIA | GLIPIZIDE |
| 146 | DRUGS USED IN DIABETES | UNCONTROLLED DIABETES<br>MELLITUS WITH<br>HYPERGLICEMIA | HUMAN MIXTARD |
| 147 | DRUGS USED IN DIABETES | UNCONTROLLED DM2 | INSULIN DETEMIR |
| 148 | UNSPECIFIED HERBAL AND TRADITIONAL MEDICINE | HERBAL SUPPLEMENT | GLYCINE MAX EXTRACT |
| 149 | LIPID MODIFYING AGENTS | DIABETES MELLITUS TYPE II | PRAVASTATIN |
| Card | liovascular (CARDDIS) | | |
| 1 | AGENTS ACTING ON THE<br>RENIN-ANGIOTENSIN SYSTEM | ACUTE MYOCARDIAL INFARCTION | IRBESARTAN |
| 2 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | CARDIOMYOPATHY | LISINOPRIL |
| 3 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | CARDIOMYOPATHY | RAMIPRIL |
| 4 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | CONGESTIVE HEART<br>FAILURE | LISINOPRIL |
| 5 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | CORONARY ARTERY DISEASE | RAMIPRIL |
| 6 | BETA BLOCKING AGENTS | ACUTE MYOCARDIAL<br>INFARCTION | BISOPROLOL FUMARATE |
| 7 | BETA BLOCKING AGENTS | ANTI-ARRHYTHMIC | SOTALOL |
| 8 | BETA BLOCKING AGENTS | ATHEROSCLEROTIC HEART<br>DISEASE OF NATIVE<br>CORONARY ARTERY<br>WITHOUT ANGINA PECTORIS | CARVEDILOL |

| | Medication Class (WHOATC2) | Indication (CMINDC) | WHOGEN |
|---|---|---|---|
| 9 | BETA BLOCKING AGENTS | ATRIAL FIBRILATION | ATENOLOL |
| 10 | BETA BLOCKING AGENTS | ATRIAL FIBRILATION | METOPROLOL |
| 11 | BETA BLOCKING AGENTS | ATRIAL FIBRILLATION | METOPROLOL |
| 12 | BETA BLOCKING AGENTS | ATRIAL FIBRILLATION | METOPROLOL TARTRATE |
| 13 | BETA BLOCKING AGENTS | ATYPICAL CHEST PAIN | LABETALOL |
| 14 | BETA BLOCKING AGENTS | BRUGADA SYNDROME | BISOPROLOL |
| 15 | BETA BLOCKING AGENTS | CAD | METOPROLOL SUCCINATE |
| 16 | BETA BLOCKING AGENTS | CADRIOMYOPATHY | BISOPROLOL |
| 17 | BETA BLOCKING AGENTS | CARDIAC PACEMAKER<br>INSITU | METOPROLOL |
| 18 | BETA BLOCKING AGENTS | CARDIAC PROPHYLAXIS | CARVEDILOL |
| 19 | BETA BLOCKING AGENTS | CARDIOMYOPATHY | CARVEDILOL |
| 20 | BETA BLOCKING AGENTS | CHEST TIGHTNESS | BISOPROLOL |
| 21 | BETA BLOCKING AGENTS | CONGESTIVE HEART<br>FAILURE | ATENOLOL |
| 22 | BETA BLOCKING AGENTS | CONGESTIVE HEART<br>FAILURE | CARVEDILOL |
| 23 | BETA BLOCKING AGENTS | CONTROLLED<br>HYPERTENSION | TENORETIC |
| 24 | BETA BLOCKING AGENTS | CORONARY ARTERY DISEASE | METOPROLOL |
| 25 | BETA BLOCKING AGENTS | CORONARY ARTERY DISEASE | METOPROLOL SUCCINATE |
| 26 | BETA BLOCKING AGENTS | CORONARY ARTERY<br>STENOSIS | METOPROLOL |
| 27 | BETA BLOCKING AGENTS | DYSRHYTHMIA | BISOPROLOL FUMARATE |
| 28 | BETA BLOCKING AGENTS | HEART FAILURE AND<br>HYPERTENSION | CARVEDILOL |
| 29 | BETA BLOCKING AGENTS | INTERMITTENT<br>ARRHYTHMIA | BISOPROLOL |
| 30 | BETA BLOCKING AGENTS | MITRAL INSUFFICIENCY | BISOPROLOL |
| 31 | BETA BLOCKING AGENTS | PREVENTATIVE FOLLOWING<br>ACUTE MYCARDIAL<br>INFARCTION | BISOPROLOL |
| 32 | BETA BLOCKING AGENTS | SICK SINUS SYNDROME | METOPROLOL |
| 33 | BETA BLOCKING AGENTS | SUPRA VENTRICULAR<br>TACHYCARDIA | ATENOLOL |
| 34 | BETA BLOCKING AGENTS | SUPRAVENTRICULAR<br>TACHYCARDIA | ATENOLOL |
| 35 | BETA BLOCKING AGENTS | SUPRAVENTRICULAR<br>TACHYCARDIA | METOPROLOL |
| 36 | BETA BLOCKING AGENTS | TACHYCARDIA | ATENOLOL |
| 37 | CALCIUM CHANNEL BLOCKERS | CORONARY ARTERY DISEASE | AMLODIPINE |
| 38 | CALCIUM CHANNEL BLOCKERS | CORONARY ARTERY DISEASE | AMLODIPINE BESILATE |
| 39 | CALCIUM CHANNEL BLOCKERS | SUPRAVENTRICULAR<br>TACHYCARDIA | VERAPAMIL |

| | Medication Class (WHOATC2) | Indication (CMINDC) | WHOGEN |
|---|---|---|---|
| 40 | CARDIAC THERAPY | ACUTE MYOCARDIAL INFARCTION | AMIODARONE HYDROCHLORIDE |
| 41 | CARDIAC THERAPY | ACUTE MYOCARDIAL INFARCTION | ISOSORBIDE DINITRATE |
| 42 | CARDIAC THERAPY | ALLERGIC REACTION | EPINEPHRINE |
| 43 | CARDIAC THERAPY | ANGINA | GLYCERYL TRINITRATE |
| 44 | CARDIAC THERAPY | ANGINA PECTORIS | RANOLAZINE |
| 45 | CARDIAC THERAPY | ANGIOGRAM/STENT | ADENOSINE |
| 46 | CARDIAC THERAPY | ANGIONEUROTIC EDEMA | EPINEPHRINE |
| 47 | CARDIAC THERAPY | ANTIARRHYTHMIC AGENT | FLECAINIDE ACETATE |
| 48 | CARDIAC THERAPY | ATRIAL FIBRILLATION | DIGOXIN |
| 49 | CARDIAC THERAPY | ATRIAL FIBRILLATION | FLECAINIDE ACETATE |
| 50 | CARDIAC THERAPY | ATYPICAL CHEST PAIN | GLYCERYL TRINITRATE |
| 51 | CARDIAC THERAPY | CAD | UBIDECARENONE |
| 52 | CARDIAC THERAPY | CARDIOMYOPATHY | ISOSORBIDE DINITRATE |
| 53 | CARDIAC THERAPY | CARDIOVASCULAR DISEASE<br>PROPHYLAXIS | UBIDECARENONE |
| 54 | CARDIAC THERAPY | CHEST PAIN | GLYCERYL TRINITRATE |
| 55 | CARDIAC THERAPY | CHEST PAINS | GLYCERYL TRINITRATE |
| 56 | CARDIAC THERAPY | CHESTPAIN | GLYCERYL TRINITRATE |
| 57 | CARDIAC THERAPY | CORONARY ARTERY DISEASE | GLYCERYL TRINITRATE |
| 58 | CARDIAC THERAPY | CORONARY ARTERY DISEASE | ISOSORBIDE MONONITRATE |
| 59 | CARDIAC THERAPY | HYPERLIPIDEMIA | ISOSORBIDE MONONITRATE |
| 60 | CARDIAC THERAPY | NSTEMI | ISOSORBIDE DINITRATE |
| 61 | CARDIAC THERAPY | PERIOP STRESS TEST | REGADENOSON |
| 62 | CARDIAC THERAPY | PROPHYLAXIS | GLYCERYL TRINITRATE |
| 63 | CARDIAC THERAPY | PROPHYLAXIS FOR CARDIAC HEALTH | UBIDECARENONE |
| 64 | CARDIAC THERAPY | SUPRAVENTRICULAR<br>TACHYCARDIA | ADENOSINE |
| 65 | CARDIAC THERAPY | UNCONTROLLED DIABETES<br>MELLITUS 2 | AMIODARONE HYDROCHLORIDE |
| 66 | CARDIAC THERAPY | UNCONTROLLED DIABETES<br>MELLITUS 2 | GLYCERYL TRINITRATE |
| 67 | DIURETICS | ACUTE RESPIRATORY<br>FAILURE | FUROSEMIDE |
| 68 | DIURETICS | AORTIC VALVE<br>REPLACEMENT | FUROSEMIDE |
| 69 | DIURETICS | CHF | BUMETANIDE |
| 70 | DIURETICS | CHF | HYDROCHLOROTHIAZIDE |
| 71 | DIURETICS | CHF | METOLAZONE |
| 72 | DIURETICS | CONGESTIVE HEART<br>FAILURE | BUMETANIDE |

| | Medication Class (WHOATC2) | Indication (CMINDC) | WHOGEN |
|---|---|---|---|
| 72 | DHIDETICG | CONGESTIVE HEART | FLIDOGEMIDE |
| 73 | DIURETICS | FAILURE | FUROSEMIDE |
| 74 | DIURETICS | CONGESTIVE HEART<br>FAILURE | HYDROCHLOROTHIAZIDE |
| 75 | DIURETICS | CONGESTIVE HEART<br>FAILURE | METOLAZONE |
| 76 | DIURETICS | CONGESTIVE HEART<br>FAILURE | SPIRONOLACTONE |
| 77 | DIURETICS | CORONARY ARTERY DISEASE | HYDROCHLOROTHIAZIDE |
| 78 | DIURETICS | CORONARY ARTERY<br>DISEASE. | FUROSEMIDE |
| 79 | DIURETICS | ELEVATION OF BLOOD<br>PRESSURE | FUROSEMIDE |
| 80 | DIURETICS | MITRAL INSUFFICIENCY | TORASEMIDE |
| 81 | DIURETICS | TRANSGENGER | SPIRONOLACTONE |
| 82 | LIPID MODIFYING AGENTS | ACUTE MYOCARDIAL INFARCTION | ATORVASTATIN CALCIUM |
| 83 | LIPID MODIFYING AGENTS | ACUTE MYOCARDIAL INFARCTION | OMEGA-3 TRIGLYCERIDES |
| 84 | LIPID MODIFYING AGENTS | ATHEROSCLEROTIC HEART<br>DISEASE OF NATIVE<br>CORONARY ARTERY<br>WITHOUT ANGINA PECTORIS | SIMVASTATIN |
| 85 | LIPID MODIFYING AGENTS | BASILAR ARTERY<br>THROMBUS | ATORVASTATIN CALCIUM |
| 86 | LIPID MODIFYING AGENTS | CAD | PRAVASTATIN SODIUM |
| 87 | LIPID MODIFYING AGENTS | CAD | ROSUVASTATIN CALCIUM |
| 88 | LIPID MODIFYING AGENTS | CARDIAC PROPHYLAXIS | ATORVASTATIN |
| 89 | LIPID MODIFYING AGENTS | CARDIAC PROPHYLAXIS | FISH OIL |
| 90 | LIPID MODIFYING AGENTS | CARDIOVASCULAR<br>PROPHYLAXIS | ATORVASTATIN CALCIUM |
| 91 | LIPID MODIFYING AGENTS | CHEST TIGHTNESS | ATORVASTATIN |
| Нур | erlipidemia (HLIPDEM) | | |
| 1 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTRIGLYCERIDEMIA | LISINOPRIL |
| 2 | ANTIHYPERTENSIVES | HYPERCHOLESTEROLEMIA | DOXAZOSIN MESILATE |
| 3 | CARDIAC THERAPY | HYPERCHOLESTEROLEMIA | UBIDECARENONE |
| 4 | LIPID MODIFYING AGENTS | ABNORMAL LIPIDS | ATORVASTATIN |
| 5 | LIPID MODIFYING AGENTS | CARDIAC PROPHYLAXIS | ROSUVASTATIN |
| 6 | LIPID MODIFYING AGENTS | CHOLESTEROL | ROSUVASTATIN |
| 7 | LIPID MODIFYING AGENTS | CHOLESTEROL | ROSUVASTATIN CALCIUM |
| 8 | LIPID MODIFYING AGENTS | CHOLESTEROLEAMIA | ATORVASTATIN |
| 9 | LIPID MODIFYING AGENTS | CHOLESTERORL | ROSUVASTATIN CALCIUM |
| 10 | LIPID MODIFYING AGENTS | CORONARY ARTERY DISEASE | ATORVASTATIN |
| 11 | LIPID MODIFYING AGENTS | CORONARY ARTERY DISEASE | EZETIMIBE |
| | Medication Class (WHOATC2) | Indication (CMINDC) | WHOGEN | |
|---|---|---|---|--|
| 12 | LIPID MODIFYING AGENTS | CORONARY ARTERY DISEASE | FENOFIBRATE | |
| 13 | LIPID MODIFYING AGENTS | CORONARY ARTERY DISEASE | ROSUVASTATIN CALCIUM | |
| 14 | LIPID MODIFYING AGENTS | CORONARY ARTERY DISEASE PROPHYLAXIS | ATORVASTATIN | |
| 15 | LIPID MODIFYING AGENTS | DIET SUPPLEMENT | FISH OIL | |
| 16 | LIPID MODIFYING AGENTS | DIETARY SUPPLEMENT | FISH OIL | |
| 17 | LIPID MODIFYING AGENTS | DIETARY SUPPLEMENTS | FISH OIL | |
| 18 | LIPID MODIFYING AGENTS | DYSLIPEDEMIA | ROSUVASTATIN CALCIUM | |
| 19 | LIPID MODIFYING AGENTS | DYSLIPIDAEMIA | ATORVASTATIN | |
| 20 | LIPID MODIFYING AGENTS | DYSLIPIDEMIA | ATORVASTATIN | |
| 21 | LIPID MODIFYING AGENTS | DYSLIPIDEMIA | FENOFIBRATE | |
| 22 | LIPID MODIFYING AGENTS | DYSLIPIDEMIA | FISH OIL | |
| 23 | LIPID MODIFYING AGENTS | DYSLIPIDEMIA | GEMFIBROZIL | |
| 24 | LIPID MODIFYING AGENTS | DYSLIPIDEMIA | PRAVASTATIN | |
| 25 | LIPID MODIFYING AGENTS | DYSLIPIDEMIA | ROSUVASTATIN | |
| 26 | LIPID MODIFYING AGENTS | DYSLIPIDEMIA, WORSENING | ROSUVASTATIN | |
| 27 | LIPID MODIFYING AGENTS | DYSLIPIDERMIA | PRAVASTATIN | |
| 28 | LIPID MODIFYING AGENTS | ELEVATED CHOLESTEROL | SIMVASTATIN | |
| 29 | LIPID MODIFYING AGENTS | ELEVATED LIPIDS | ATORVASTATIN | |
| 30 | LIPID MODIFYING AGENTS | ELEVATED LIPIDS | ATORVASTATIN CALCIUM | |
| 31 | LIPID MODIFYING AGENTS | ELEVATED TRIGLYCERIDES | FISH OIL | |
| 32 | LIPID MODIFYING AGENTS | HIGH CHOLESTEROL | ATORVASTATIN | |
| 33 | LIPID MODIFYING AGENTS | HIGH CHOLESTEROL | ATORVASTATIN CALCIUM | |
| 34 | LIPID MODIFYING AGENTS | HIGH CHOLESTEROL | GEMFIBROZIL | |
| 35 | LIPID MODIFYING AGENTS | HIGH CHOLESTEROL | LOVASTATIN | |
| 36 | LIPID MODIFYING AGENTS | HIGH CHOLESTEROL | PRAVASTATIN | |
| 37 | LIPID MODIFYING AGENTS | HIGH CHOLESTEROL | ROSUVASTATIN CALCIUM | |
| 38 | LIPID MODIFYING AGENTS | HIGH CHOLESTEROL | SIMVASTATIN | |
| 39 | LIPID MODIFYING AGENTS | HIGH CHOLESTROL | ATORVASTATIN | |
| 40 | LIPID MODIFYING AGENTS | HIGH PLASMA LIPIDS | ATORVASTATIN | |
| 41 | LIPID MODIFYING AGENTS | HIGH TRIGLYCERIDES | FENOFIBRATE | |
| 42 | LIPID MODIFYING AGENTS | HIGH TRIGLYCERIDES AND<br>HYPERCHOLESTEROLEMIA | ATORVASTATIN | |
| 43 | LIPID MODIFYING AGENTS | HIPERCOLESTEROLEMIA | ATORVASTATIN | |
| 44 | LIPID MODIFYING AGENTS | HIPERCOLESTEROLEMIA | ATORVASTATIN CALCIUM | |
| 45 | LIPID MODIFYING AGENTS | HIPERCOLESTEROLEMIA | SIMVASTATIN | |
| 46 | LIPID MODIFYING AGENTS | HYERLIPIDEMIA | OMEGA-3-ACID ETHYL ESTER | |
| 47 | LIPID MODIFYING AGENTS | HYPERCHOLESTERIMIA | FENOFIBRATE | |
| 48 | LIPID MODIFYING AGENTS | HYPERCHOLESTERINAEMIA | ATORVASTATIN | |
| 49 | LIPID MODIFYING AGENTS | HYPERCHOLESTERINAEMIA | PRAVASTATIN | |
| 50 | LIPID MODIFYING AGENTS | HYPERCHOLESTERINEMIA | PRAVASTATIN | |
| 51 | LIPID MODIFYING AGENTS | HYPERCHOLESTERINEMIA | SIMVASTATIN | |

| | Medication Class (WHOATC2) | Indication (CMINDC) | WHOGEN |
|---|---|---|---|
| 52 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROL | PRAVASTATIN |
| 53 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROLAEMIA | ATORVASTATIN |
| 54 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROLAEMIA | PRAVASTATIN |
| 55 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROLAEMIA | ROSUVASTATIN |
| 56 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROLAEMIA | SIMVASTATIN |
| 57 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROLEMIA | ATORVASTATIN |
| 58 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROLEMIA | ATORVASTATIN CALCIUM |
| 59 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROLEMIA | EZETIMIBE |
| 60 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROLEMIA | FENOFIBRATE |
| 61 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROLEMIA | FISH OIL |
| 62 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROLEMIA | LOVASTATIN |
| 63 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROLEMIA | PITAVASTATIN CALCIUM |
| 64 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROLEMIA | PRAVASTATIN |
| 65 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROLEMIA | PRAVASTATIN SODIUM |
| 66 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROLEMIA | ROSUVASTATIN |
| 67 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROLEMIA | ROSUVASTATIN CALCIUM |
| 68 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROLEMIA | SIMVASTATIN |
| 69 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROLEMIA<br>(PURE) AND MIXED<br>HYPERLIPIDEMIA | ROSUVASTATIN CALCIUM |
| 70 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROLMIA | PRAVASTATIN SODIUM |
| 71 | LIPID MODIFYING AGENTS | HYPERCHOLESTROLEMIA | ATORVASTATIN |
| 72 | LIPID MODIFYING AGENTS | HYPERCHOLESTROLEMIA | ATORVASTATIN CALCIUM |
| 73 | LIPID MODIFYING AGENTS | HYPERCHOLESTROLEMIA | FENOFIBRATE |
| 74 | LIPID MODIFYING AGENTS | HYPERCHOLSTEROAEMIA | ATORVASTATIN CALCIUM |
| 75 | LIPID MODIFYING AGENTS | HYPERCOLESTEROLEMIA | SIMVASTATIN |
| 76 | LIPID MODIFYING AGENTS | HYPERLIDEMIA | ROSUVASTATIN CALCIUM |
| 77 | LIPID MODIFYING AGENTS | HYPERLIDIPEMIA | ATORVASTATIN |
| 78 | LIPID MODIFYING AGENTS | HYPERLIPDEMIA | ROSUVASTATIN CALCIUM |
| 79 | LIPID MODIFYING AGENTS | HYPERLIPEDMIA-MIXED | ATORVASTATIN |
| 80 | LIPID MODIFYING AGENTS | HYPERLIPIDAEMIA | ATORVASTATIN |
| 81 | LIPID MODIFYING AGENTS | HYPERLIPIDAEMIA | FENOFIBRATE |
| 82 | LIPID MODIFYING AGENTS | HYPERLIPIDAEMIA | PRAVASTATIN |
| 83 | LIPID MODIFYING AGENTS | HYPERLIPIDAEMIA | PRAVASTATIN SODIUM |
| 84 | LIPID MODIFYING AGENTS | HYPERLIPIDAEMIA | ROSUVASTATIN |
| 85 | LIPID MODIFYING AGENTS | HYPERLIPIDAEMIA | ROSUVASTATIN CALCIUM |
| 86 | LIPID MODIFYING AGENTS | HYPERLIPIDEMA | ATORVASTATIN |
| 87 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA | ATORVASTATIN |
| 88 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA | ATORVASTATIN CALCIUM |
| 89 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA | COLESEVELAM HYDROCHLORIDE |
| 90 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA | EICOSAPENTAENOIC ACID ETHYL ESTER |

| | Medication Class (WHOATC2) | Indication (CMINDC) | WHOGEN |
|---|---|---|---|
| 91 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA | EZETIMIBE |
| 92 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA | FENOFIBRATE |
| 93 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA | FENOFIBRIC ACID |
| 94 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA | FISH OIL |
| 95 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA | GEMFIBROZIL |
| 96 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA | LOVASTATIN |
| 97 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA | OMEGA-3-ACID ETHYL ESTER |
| 98 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA | PELAGO |
| 99 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA | PRAVASTATIN |
| 100 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA | PRAVASTATIN SODIUM |
| 101 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA | ROSUVASTATIN |
| 102 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA | ROSUVASTATIN CALCIUM |
| 103 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA | SIMVASTATIN |
| 104 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA<br>PREVENTION | ROSUVASTATIN CALCIUM |
| 105 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA, | PRAVASTATIN |
| 106 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA, MIXED | ATORVASTATIN CALCIUM |
| 107 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA, MIXED | FENOFIBRATE |
| 108 | LIPID MODIFYING AGENTS | HYPERTENSION | ATORVASTATIN |
| 109 | LIPID MODIFYING AGENTS | HYPERTENSION | PRAVASTATIN |
| 110 | LIPID MODIFYING AGENTS | HYPERTRIGLYCERDEMIA | ATORVASTATIN |
| 111 | LIPID MODIFYING AGENTS | HYPERTRIGLYCERIDEMIA | ATORVASTATIN CALCIUM |
| 112 | LIPID MODIFYING AGENTS | HYPERTRIGLYCERIDEMIA | FENOFIBRATE |
| 113 | LIPID MODIFYING AGENTS | HYPERTRIGLYCERIDEMIA | FENOFIBRIC ACID |
| 114 | LIPID MODIFYING AGENTS | HYPERTRIGLYCERIDEMIA | FIBRATES |
| 115 | LIPID MODIFYING AGENTS | HYPERTRIGLYCERIDEMIA | FISH OIL |
| 116 | LIPID MODIFYING AGENTS | HYPERTRIGLYCERIDEMIA | OMEGA-3 TRIGLYCERIDES |
| 117 | LIPID MODIFYING AGENTS | HYPERTRIGLYCERIDEMIA | PRAVASTATIN |
| 118 | LIPID MODIFYING AGENTS | HYPERTRIGLYCERIDEMIA,HY<br>PERCHOLESTEROLEMIA | ATORVASTATIN |
| 119 | LIPID MODIFYING AGENTS | HYPERTRIGLYERIDEMIA | GEMFIBROZIL |
| 120 | LIPID MODIFYING AGENTS | HYPERTRYGLYCERIDEMIA | PRAVASTATIN |
| 121 | LIPID MODIFYING AGENTS | INDICATION<br>HYPERLIPIDEMIA | FENOFIBRATE |
| 122 | LIPID MODIFYING AGENTS | IRRITABLE BOWEL<br>SYNDROME | FISH OIL |
| 123 | LIPID MODIFYING AGENTS | ISCHEMIC HEART DISEASE | ROSUVASTATIN CALCIUM |
| 124 | LIPID MODIFYING AGENTS | LDL-CHOLESTEROL GRADE 3<br>ELEVATION | ROSUVASTATIN |
| 125 | LIPID MODIFYING AGENTS | MIXED DYSLIPIDEMIA | FENOFIBRATE |
| 126 | LIPID MODIFYING AGENTS | MIXED DYSLIPIDEMIA | ROSUVASTATIN CALCIUM |
| 127 | LIPID MODIFYING AGENTS | MIXED HYPERLIPDEMIA | ATORVASTATIN |

| | Medication Class (WHOATC2) | Indication (CMINDC) | WHOGEN |
|---|---|---|---|
| 128 | LIPID MODIFYING AGENTS | MIXED HYPERLIPIDEMIA | ATORVASTATIN |
| 129 | LIPID MODIFYING AGENTS | MIXED HYPERLIPIDEMIA | FENOFIBRATE |
| 130 | LIPID MODIFYING AGENTS | MIXED HYPERLIPIDEMIA | GEMFIBROZIL |
| 131 | LIPID MODIFYING AGENTS | NUTRITION SUPPLEMENT | FISH OIL |
| 132 | LIPID MODIFYING AGENTS | NUTRITIONAL SUPPLEMENT | FISH OIL |
| 133 | LIPID MODIFYING AGENTS | NUTRITIONAL SUPPLEMENT | OMEGA-3 FATTY ACIDS |
| 134 | LIPID MODIFYING AGENTS | PREVENTATIVE FOLLOWING<br>ACUTE MYCARDIAL<br>INFARCTION | ATORVASTATIN |
| 135 | LIPID MODIFYING AGENTS | PREVENTION FOR<br>HYPERCHOLESTEROLEMIA | OMEGA-3 FATTY ACIDS |
| 136 | LIPID MODIFYING AGENTS | PREVENTIVE | FISH OIL W/LINUM<br>USITATISSIMUM SEED OIL |
| 137 | LIPID MODIFYING AGENTS | PROPHYLAXIS | FISH OIL |
| 138 | LIPID MODIFYING AGENTS | PURE<br>HYPERCHOLESTEROLEMIA | ATORVASTATIN |
| 139 | LIPID MODIFYING AGENTS | SECONDARY STROKE<br>PREVENTION | ATORVASTATIN |
| 140 | LIPID MODIFYING AGENTS | STROKE PROPHYLAXIS | ATORVASTATIN |
| 141 | LIPID MODIFYING AGENTS | SUPPLEMENT | FISH OIL |
| 142 | LIPID MODIFYING AGENTS | SUPPLEMENT | OMEGA 3 6 9 |
| 143 | LIPID MODIFYING AGENTS | SUPPLEMENT | OMEGA-3 FATTY ACIDS |
| 144 | LIPID MODIFYING AGENTS | SUPPLEMENT | OMEGA-3 FATTY ACIDS W/OMEGA-6 FATTY ACIDS |
| 145 | LIPID MODIFYING AGENTS | SUPPLEMENT | OMEGA-3-ACID ETHYL ESTER |
| 146 | LIPID MODIFYING AGENTS | SUPPLEMENT/HYPERLIPIDEM IA | FISH OIL |
| 147 | LIPID MODIFYING AGENTS | SUPPLEMENTAL USE | FISH OIL |
| 148 | LIPID MODIFYING AGENTS | SUPPLEMETN | FISH OIL |
| 149 | LIPID MODIFYING AGENTS | UNCONTROLLED DIABETES<br>MELLITUS 2 | ATORVASTATIN |
| 150 | LIPID MODIFYING AGENTS | WORSENING<br>HYPERLIPIDEMIA | ATORVASTATIN |
| 151 | LIPID MODIFYING AGENTS | WORSENING OF<br>HYPERLIPIDEMIA | FISH OIL |
| 152 | LIPID MODIFYING AGENTS | HIGH CHOLESTEROL | NICOTINIC ACID |
| 153 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROLEMIA | NICOTINIC ACID |
| 154 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA | NICOTINIC ACID |
| 155 | LIPID MODIFYING AGENTS | MIXED HYPERLIPIDEMIA | NICOTINIC ACID |

# **Appendix 4.** Hepatic Events

An adverse event record will be flagged as a hepatic event if its MedDRA PT included in the pre-specified PT list, which includes all PTs from the broad search of the following 15 SMQs under MedDRA 19.1 provided by Gilead DSPH and reviewed by Gilead medical monitors.

| | SMQ Source |
|---|---|
| Hepatic Events (HEP) | Biliary neoplasms benign (incl cysts and polyps) (SMQ) |
| | Biliary malignant tumours (SMQ) |
| | Biliary tumours of unspecified malignancy (SMQ) |
| | Biliary system related investigations, signs and symptoms (SMQ) |
| | Biliary tract disorders (SMQ) |
| | Gallbladder related disorders (SMQ) |
| | Gallstone related disorders (SMQ) |
| | Cholestasis and jaundice of hepatic origin (SMQ) |
| | Hepatic failure, fibrosis and cirrhosis and other liver damage-related conditions (SMQ) |
| | Hepatitis, non-infectious (SMQ) |
| | Liver neoplasms, benign (incl cysts and polyps) (SMQ) |
| | Liver malignant tumours (SMQ) |
| | Liver tumours of unspecified malignancy (SMQ) |
| | Liver related investigations, signs and symptoms (SMQ) |
| | Liver-related coagulation and bleeding disturbances (SMQ) |

## **Appendix 5. Programming Specification**

- 1. AGE calculated as follows:
  - a. AGE (years) is calculated from the number of days between the date of birth (DOB) and Day 1 (randomized phase first dose date),
  - b. Use the SAS INTCK function to determine the number of "1st-of-month days" (eg, January 1st, February 1st, March 1st) between DOB and Day 1 (inclusive),
  - c. Divide the result in (b) by 12,
  - d. AGE = the integer of the result in (c),
  - e. If the DOB and randomized phase Day 1 have the month in common and the birthday is later in the month than the date of randomized phase Study Day 1, then subtract one from the AGE result above.

For subjects randomized and never dosed with study drug, age will be calculated from the date of randomization

- 2. All screened subjects refer to all subjects who are screened (ie, with nonmissing screening date) and have a screening number. For summaries, the same subject is counted only once. DOB and other demographic information such as sex, race, ethnicity, country, and initials will be used to identify unique screened subjects.
- 3. Screen failure subjects are the subjects who are screened and answered "No" for any inclusion criteria or "Yes" for any exclusion criteria regardless of which version of protocol the subject was consent to.
- 4. Subjects in the randomized analysis set are defined as subjects randomized into the study. IXRSRAND is the source to determine whether the subject is randomized (ie, subject with nonmissing RGMNDTN in the IXRSRAND dataset) and confirmed by the eCRF ENROLL dataset (ie, ENROLLYN = "Yes" in ENROLL dataset).
- 5. Randomized treatment (ie, TRT01P in ADSL) are derived from IXRSRAND, while actual treatment received (ie, TRT01A in ADSL) is assigned as the randomized treatment if subject took at least 1 dose of randomized study drug and assigned as blank if subject never dosed.
- 6. In disposition table, the reasons for premature discontinuation are displayed in the order as they appear on the eCRF.
- 7. Only 1 study completion form is collected for the entire study. Therefore, study disposition in the randomized phase of the study is defined as follows for subjects who were dosed with randomized study drug:

- a) Subjects who completed study in the randomized phase include the following two exclusive cases:
  - i) Subjects who were dosed in the extension phase (ie, extension phase first dose date is present), OR
  - ii) Subjects who were not dosed in the extension phase and completed study (ie, extension phase first dose date is not present and study completion form is marked as "Yes")
- b) Subjects who are ongoing in the randomized phase of the study include subjects who were not dosed in the extension phase of the study, and study completion form was not filled.
- c) Subjects who discontinued study in the randomized phase of the study include subjects who were not dosed in the extension phase of the study and study completion form was marked as "No".
- 8. Body mass index (BMI) and Body Surface Area (BSA)

BMI and BSA will be calculated only at randomized phase baseline as follows:

```
    BMI = (weight [kg])/ (height [meters]<sup>2</sup>)
    BSA (m<sup>2</sup>) = SQRT( [Height(cm) x Weight(kg) ]/ 3600 )
```

Baseline height and weight in the randomized phase of the study will be used for this calculation.

- 9. SAS codes for the treatment comparison for demographics and baseline characteristics tables.
  - 1) CMH test for nominal variable (Y), the p-value from general association test should be used for nominal variable:

```
proc freq order=adsl;
   tables trtgrp * Y /cmh /*general association test*/
run;
```

2) CMH test for ordinal variable (Y), the p-value from row mean score test should be used for ordinal variable:

```
proc freq order=adsl;
   tables trtgrp * Y / cmh2 ; /*row mean score test*/
run;
```

3) Wilcoxon rank sum test for continuous variable (Y), the p-value from the normal approximation two-sided test should be used for continuous variable:

```
proc npar1way wilcoxon data=adsl;
    class trtgrp;
    var Y;
run;
```

Note: "Not Permitted", "Unknown", or missing categories will be excluded for percentage calculation and also be excluded for p-value generation for categorical data analysis (eg, CMH test or Fisher exact test), except for Mode of Infection (HIV Risk Factors), where "Unknown" will be included for percentage calculation since a subject may fit more than 1 HIV risk factors. For this variable, percentage may add up to be more than 100% and no p-value will be generated.

Subjects with Race = "Not Permitted" will also be excluded to define Race subgroup (ie, back vs. nonblack) for efficacy subgroup analysis.

10. SAS code for the treatment comparison for duration of exposure. The p-value from log rank test should be used.

- 11. Last Dose Date and Last Study Date
  - 1) Last Dose Date (ie, TR01EDTC and TR01EDT for randomized phase last dose date, and TR02EDTC and TR02EDT for extension phase last dose date) in ADSL was defined in Section 3.8.1.

#### Randomized Phase Last Dose Date:

For subjects with a partial last dosing date (ie, month and year of last dose are known), the minimum of {(death date, if available), (extension phase first dose date – 1 day, if available), (the latest of the dispensing dates of study drug bottles, study drug start dates and end dates (based on EX dataset), and the imputed last dose date [day imputed as 15])} will be used as the final imputed last dose date. However if dispensing date's month is after last dose date's month, data query is needed.

Please note the follows:

• Last dose date is not defined for subjects still on randomized study drug. However, for the calculation of the duration of exposure to randomized study drug, the data cut date will be used to impute the last dose date for subjects who have not discontinued study drug by the data cut date. For Week 48 interim analysis, 22 Sep 2017 will be the data cut date for subjects with Week 48 visit on or prior to 22 Sep 2017, subjects missing Week 48 visits while on study drug, or subjects who permanently discontinued the

randomized study drug. For subjects with Week 48 visit after 22 Sep 2017, the last subject's Week 48 visit date will be used as the data cut date.

For time to premature discontinuation of study drug KM summary, if we have subjects with duration of exposure of study drug great than 378 days (ie, upper limit of the Week 48 visit window), please add Week 60, defined as Day 379 – Day 462 (inclusive), to the table.

#### **Extension Phase Last Dose Date:**

For subjects with a partial last dosing date (ie, month and year of last dose are known), the minimum of {(death date, if available), (the latest of the dispensing dates of study drug bottles, study drug start dates and end dates (based on EX dataset), and the imputed last dose date [day imputed as 15])} will be used as the final imputed last dose date. However if dispensing date's month is after last dose date's month, data query is needed.

Last dose date is not defined for subjects still on study drug in SAP. However, for programing purposes, the data cut date will be used to impute the last dose date for subjects still on study drug.

2) Last Study Date is the latest of the study drug start dates and end dates, the clinic visit dates, and the laboratory visit dates, including the 30-day follow-up visit date, for subjects who prematurely discontinued study or who completed study according to the Study Completion eCRF. If study drug start dates or end dates is partially missing (ie, only year and month are known), the day will be imputed as 15 for the purpose of this analysis.

Last study date is not defined for subjects still on study in SAP. However, for programing purpose, the latest of data cut date, the clinic visit dates, and the laboratory visit dates, including the 30-day follow-up visit date, will be used to impute the last study date for subjects still on study.

#### 12. Toxicity Grades:

- 1) For toxicity grade summaries, include all postbaseline graded results up to 30 days after the randomized phase last dose of study drug, not just those used in by-visit summaries
- 2) For glucose grading, as specified in SAP Section 7.2.2.1, the treatment-emergent flag cannot be determined for nonfasting glucose (including glucose results without a known fasting status). As a result, these records will be excluded from the "Maximum Treatment-emergent Toxicity Grade" summary in the "Treatment-emergent Laboratory Abnormalities" or "Treatment-emergent Grade 3 or 4 Laboratory Abnormalities" summary tables. In addition, fasting glucose and non-fasting glucose will be listed as two separate laboratory tests in the "Laboratory Abnormalities" and

"Grade 3 or 4 Laboratory Abnormalities" listings. Only a maximum postbaseline toxicity flag will be displayed and the treatment-emergent flag will not be displayed for nonfasting glucose as the treatment-emergent flag cannot be determined for nonfasting glucose.

## 13. Efficacy analyses:

1) For categorical efficacy response (eg, Subjects with HIV-1 RNA ≥ 50 copies/mL or Subjects with HIV-1 RNA < 50 copies/mL as determined by US FDA-defined snapshot algorithm, M=F or M=E Analyses): the proportion difference between 2 treatment groups and its 95.001% CIs (or 95% CI for M=F and M=E analyses) are calculated based on the an unconditional exact method with 2 inverted 1-sided tests in SAS v9.3 or above. Please see example SAS codes below:

```
data example;
input grp trt01a $ outcome $ count ;
datalines;

      1
      Treat-A
      2-Fail

      1
      Treat-A
      1-Succ

      1
      Treat-B
      2-Fail

      1
      Treat-B
      1-Succ

                                               1
                                            189
                                              4
                                             88
run;
proc freq data = example;
table trt01a*outcome /riskdiff(CL=(exact)) alpha=0.04999;
weight count; exact RISKDIFF(METHOD=SCORE);
output out=ciexact(keep= RDIF1 XL RDIF1 XU RDIF1) riskdiff;
data final(keep=A1 B1 Estimate LowerCL UpperCL ocharcl);
set ciexact;
label Estimate ="Percentage Difference"
LowerCL = "95% Lower Confidence Limit"
UpperCL = "95% Upper Confidence Limit"
A1 = "Percentage of Success in Treat-A"
B1 = "Percentage of Success in Treat-B";
Estimate=100* RDIF1 ;
LowerCL = 100*XL RDIF1;
UpperCL = 100*XU RDIF1;
A1 = 100* RSK11 ;
B1 = 100* RSK21;
ocharc1 = right(compress(put(Estimate, 8.1)) || '% (' ||
compress(put(LowerCL, 8.1)) || '% to ' || compress(put(UpperCL, 8.1)) || '%)');
run;
```

2) Homogeneity test: Homogeneity Test of Treatment Effect across country in HIV-1 RNA < 50 copies/mL at Week 48 (Snapshot Algorithm). For each country, the odds ratio and its 95% CI are calculated from the CMH test. For overall, the odds ratio and its 95% CI are calculated based on the common odds ratio estimate from the CMH test. The p-value for the homogeneity test is based on the Breslow-Day test of the interaction between country and treatment group as follows.

```
proc freq data=xxx;
    tables country*treat*Y/all; /*p value from Breslow Day test*/
run;
```

3) Homogeneity test: Homogeneity Test of Treatment Effect between Subgroups in HIV-1 RNA < 50 copies/mL at Week 48 (Snapshot Algorithm)

For the subgroups of age, race, and region (US vs. Ex-US) the odds ratio and the associated 95% CIs are estimated for the response variable (response coded as 1 for success and 0 for nonsuccess) using a logistic regression model including treatment (trtgrp coded as 1 for active [ie, B/F/TAF] and 2 for control [ie, SBR]), subgroup factor (coded as 1 for the first subgroup and 2 for the second subgroup), and treatment by subgroup factor. For example, for the age subgroup (agegrp coded as 1 for < 50 and 2 for  $\ge$  50), the following SAS code will be used to generate the Odds Ratio and its 95% CI within the subgroup:

Note: For the following code, it is assumed that none of the variables have any formats applied to them. If they do, they must be removed before calling the code.

```
proc genmod data=data descending;
  class trtgrpn agegrp;
  model response = trtgrpn agegrp trtgrpn*agegrp/dist=bin
  link=logit lrci;
  estimate 'Group 1' trtgrpn 1 -1 trtgrpn*agegrp 1 0 -1 0/exp;
  estimate 'Group 2' trtgrpn 1 -1 trtgrpn*agegrp 0 1 0 -1/exp;
run;
```

Note: P-value for the homogeneity test was based on the Wald test of the interaction between treatment and subgroup. Odds ratio is from L'Beta estimate, its 95%CI is from L'Beta confidence limits for each subgroup.

4) ANOVA model for continuous efficacy variable (eg, CD4+): The differences in changes from baseline in CD4+ cell count between treatment groups and the associated 95% CI will be constructed using an ANOVA, including treatment as fixed effects in the model.

```
proc glm data=adeff;
     class trtgrp;
     model CD4= trtgrp;
     lsmeans trtgrp /alpha=0.05 cl pdiff;
run;
```

5) Listing for US FDA-defined snapshot outcome:

In addition to flagging the values of HIV-1 RNA < 50 or  $\ge 50$  copies/mL for virologic outcomes, flag the last available HIV-1 RNA value while on treatment for the following categories:

- a. HIV-1 RNA >= 50 copies/mL Discontinued Study Drug Due to AE or Death and Last Available HIV-1 RNA >= 50 copies/mL
- b. HIV-1 RNA >= 50 copies/mL Discontinued Study Drug Due to Other reason\* and Last Available HIV-1 RNA >= 50 copies/mL
- c. No virologic Data Discontinued Study Drug Due to AE or Death and Last Available HIV-1 RNA < 50 copies/mL
- d. No virologic Data Discontinued Study Drug Due to Other reason\* and Last Available HIV-1 RNA < 50 copies/mL

Note: \*Other reasons include subjects who discontinued study drug due to investigator's discretion, subject decision, lost to follow-up, noncompliance with study drug, protocol violation, pregnancy, and study terminated by sponsor.

- 6) Snapshot definition clarification:
  - a. For a subject who completed the randomized phase study with Week 48 HIV-1 RNA missing for the randomized phase of the study, snapshot outcome for such subject would be "Missing data during the window but on study drug".
- 14. Clarification of the LOCF algorithms for CD4: (1) baseline value will be carried forward; (2) if a value is missing in an analysis visit window, replace the missing value with the last on-treatment value observed before the analysis visit window that has the missing value.
- 15. Graded Laboratory Abnormalities Summary

The following labels will be used for treatment-emergent laboratory abnormalities and treatment-emergent Grade 3 or 4 laboratory abnormalities summary tables and listings:

| Battery | Lab Test Label<br>Used in l-labtox Listing | Toxicity<br>Direction | Lab Test Label Used in t-labtox Table |
|---|---|---|---|
| Hematology | Hemoglobin | Decrease | Hemoglobin (Decreased) |
| | Neutrophils | Decrease | Neutrophils (Decreased) |
| | Platelets | Decrease | Platelets (Decreased) |
| | WBC | Decrease | WBC (Decreased) |
| Chemistry | Albumin | Decrease | Albumin (Decreased) |
| | Alkaline Phosphatase | Increase | Alkaline Phosphatase (Increased) |
| | ALT | Increase | ALT (Increased) |
| | Amylase | Increase | Amylase (Increased) |
| | AST | Increase | AST (Increased) |
| | Bicarbonate | Decrease | Bicarbonate (Decreased) |
| | Corrected Calcium | Increase | Corrected Calcium (Hypercalcemia) |
| | Corrected Calcium | Decrease | Corrected Calcium (Hypocalcemia) |
| | Creatine Kinase (CK) | Increase | Creatine Kinase (Increased) |
| | Creatinine | Increase | Creatinine (Increased) |
| | GGT | Increase | GGT (Increased) |
| | Lipase | Increase | Lipase (Increased) |
| | Magnesium | Decrease | Magnesium (Hypomagnesemia) |
| | Phosphate | Decrease | Phosphate (Hypophosphatemia) |
| | Serum Glucose (Fasting) | Increase | Serum Glucose (Fasting, Hyperglycemia) |
| | Serum Glucose (Fasting) | Decrease | Serum Glucose (Fasting, Hypoglycemia) |
| | Serum Glucose (Nonfasting) | Increase | Serum Glucose (Nonfasting, Hyperglycemia) |
| | Serum Glucose (Nonfasting) | Decrease | Serum Glucose (Nonfasting, Hypoglycemia) |
| | Serum Potassium | Increase | Serum Potassium (Hyperkalemia) |
| | Serum Potassium | Decrease | Serum Potassium (Hypokalemia) |
| | Serum Sodium | Increase | Serum Sodium (Hypernatremia) |
| | Serum Sodium | Decrease | Serum Sodium (Hyponatremia) |
| | Total Bilirubin | Increase | Total Bilirubin (Hyperbilirubinemia) |
| | Total Cholesterol (Fasting) | Increase | Total Cholesterol (Fasting, Hypercholesterolemia) |
| | Triglycerides (Fasting) | Increase | Triglycerides (Fasting, Increased) |
| | LDL (Fasting) | Increase | LDL (Fasting, Increased) |
| | Urea Nitrogen (BUN) | Increase | Urea Nitrogen (Increased) |
| | Uric Acid | Increase | Uric Acid (Hyperuricemia) |

| Battery | Lab Test Label<br>Used in l-labtox Listing | Toxicity<br>Direction | Lab Test Label Used in t-labtox Table |
|---|---|---|---|
| | Uric Acid | Decrease | Uric Acid (Hypouricemia) |
| | Prothrombin Intl.<br>Normalized Ratio (INR) | Increase | N/A |
| | Prothrombin Time (PT) | Increase | N/A |
| Urinalysis | Urine Blood | Increase | N/A |
| | Urine Glucose | Increase | Urine Glucose (Glycosuria) |
| | Urine Protein | Increase | Urine Protein (Proteinuria) |
| | Urine RBC | Increase | Urine RBC (Hematuria, Quantitative) |

Note: Prothrombin Intl. Normalized Ratio (INR) and Prothrombin Time (PT) were graded based on the protocol defined toxicity grade scale. The results and toxicity grade will be listed in listing, but not be summarized in lab toxicity summary table.

## 16. Renal related laboratory evaluation

- 1) Unit conversion for renal safety tests derived from related tests with conventional units
  - a) Urine RBP (ug/L) to creatinine (mg/dL) ratio:  $1 (ug/L) / (mg/dL) = 100 \times ug/g$
  - b) Urine Beta-2-microglobulin (mg/L) to creatinine (mg/dL) ratio:  $1 \text{ (mg/L)} / \text{ (mg/dL)} = 10^5 \text{ ug/g}$
  - c) Urine Albumin (mg/dL) to creatinine (mg/dL) ratio: 1 (mg/dL) / (mg/dL) = 1000 x mg/g

#### 2) Calculation of ratios:

To calculate laboratory ratios (eg, urine RBP to creatinine ratio), the lab value of each test in the ratio needs to be from the same accession number; if any test value used for the ratio calculation from the same accession number is missing, then the ratio is not calculable (ie, missing).

### 17. Smoking history at baseline

Smoking history at baseline (ie, never smoker, former smoker, and current smoker) will be summarized as part of the baseline disease characteristics. How to classify a subject as never, former, or current smoker is specified as follows:

- a. First, select only records with *Type of Substance Use* = "Cigarettes" or "Cigars". Records with *Type of Substance Use* = "Other" (including chew tobacco, e-cigarettes, etc) will not be considered as smoking.
- b. Second, for each selected substance use record, flag whether it is "Prior", "Present", or "Post" relative to the first dose date according to the Algorithm below.

c. Finally, the subject will be flagged as "Never smoker", if the subject has no record with *Type of Substance Use* = "Cigarettes" or "Cigars" or all selected records have a flag of "Post"; the subject will be flagged as a "Former" smoker, if all selected records have a flag of "Prior" or a combination of "Prior" and "Post"; Otherwise, the subject will be flagged as a "Current" smoker.

| | | Selected Substance Use Records | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Prior | No | No | Yes | Yes | Yes | No | No | Yes |
| Present | No | No | No | No | Yes | Yes | Yes | Yes |
| Post | No | Yes | No | Yes | No | No | Yes | Yes |
| Smoking History | Never | Never | Former | Former | Current | Current | Current | Current |

# Algorithm to flag whether a selected record is "Prior", "Present", or "Post" relative to the first dose date:

- The start and stop dates of the selected record are not missing (ie, at least year is known) or the start date is not missing and record is ongoing. The completed start or stop dates will be used to compare with the first dose date whenever possible.
   Otherwise, the month and year (or year alone if month is not recorded) of the start or stop dates will be used to compare with the first dose date when the start or stop date of the selected record is incomplete.
  - a. The record is flagged as "Prior", if the stop date is before (<) the first dose date;
  - b. The record is flagged as "Present", if the start date is on or before (≤) the first dose date and the stop date is on or after (≥) the first dose date, or the selected record is marked as ongoing and the start date is on or before (≤) the first dose date:
  - c. The record is flagged as "Post", if the start date is after the first dose date;
- 2. The start date of the selected record is completely missing. We assume that the start date is before the first dose date, the stop date (or the month and/or year of the stop date, if stop date is incomplete) will be used to determine whether the selected record is "Prior" or "Present" as follows.
  - a. The record is flagged as "Prior", if the stop date is before (<) the first dose date or the stop date is completed missing and the record is not marked as ongoing.
  - b. The record is flagged as "Present", if the stop date is on or after (≥) the first dose date or the selected record is marked as ongoing.
- 3. The start date of the selected record is before (<) the first dose date, but the stop date is completely missing and the record is not marked as ongoing. We assume that the end date is before the first dose date, the record is flagged as "Prior".

4. The start date of the selected record is on or after the first dose date, but the stop date is completely missing and the record is not marked as ongoing. This is a data issue and should be queried first. However, this record is flagged as "Present" if the start date is on the first dose date; this record is flagged as "Post" if the start date is after the first dose date.

Note: first dose date for smoking history definition at baseline refers to the randomized phase first dose date.

- 18. Clarification for "Pharmacokinetic Blood Sampling Time Record" listing
  - A new variable "Sample age" will be added in this listing, defined as the duration in day between sample collection date and assay date, ie, sample age = assay date sample collection date + 1.
  - SAMTIME (hours) = sample collection time (xx:xx) last dose time before sample collection (xx:xx).
- 19. Non-study drug ARV medications (ie, ARV medications other than study drug that are taken while receiving study drug) will be flagged in "Antiviral Medication" listing. Please note that for ARVs recorded on the "Prior ARV" eCRF will NOT be considered as ARVs taken during study. All Prior ARVs with missing end date will be queried to confirm the ARVs were stopped before the randomized phase 1<sup>st</sup> dose date.
- 20. Lipid modifying medication analyses:
  - Lipid modifying medication is defined to be the concomitant medication with CMCLAS = "LIPID MODIFYING AGENTS" and CMDECOD contains wording of "STATIN" in the ADCM dataset.
  - Subjects who took lipid modifying medications at study entry refer to the subjects who use of the lipid modifying agents at study day 1 (ie, the randomized phase first dose date). More specifically, subjects with "Lipid Modifying Agent Use at Study Entry" include those subjects in safety analysis set with: 1) any selected CM record with the start date ≤ the randomized phase first dose date, and 2) the end date of the selected CM record is ongoing or the end date of the selected CM record ≥ the randomized phase first dose date.
  - Subjects who initiated lipid modifying medications during the randomized phase study include the following subjects in the safety analysis set: (1) for subjects who permanently discontinued randomized phase study drug with any selected CM record started after the randomized phase first dose date and on and prior to the minimum of randomized phase last dose date and (extension phase first dose date minus 1 day); (2) for subjects who are still on randomized study drug (if applicable) with any selected CM records started after the randomized phase first dose date; (3) lastly, for subjects who meet criteria (1) or (2) above, if they took lipid modification medications at study entry, they will be NOT be considered taking lipid modifications during the randomized phase study.

- For lipid modifying medications with start date completely unknown, we assume the start date is on or before the randomized phase first dose date, lipid modifying medication was considered as being taken at study entry if the end date is not prior to the first dose date (ie, the end date is on or after the first dose date, completely unknown, or ongoing).
- Lipid modifying medications with the start date on or prior to the randomized phase first
  dose date and the end date completely unknown were considered as being taken at study
  entry.
- 21. For figures, if at a visit where n (sample size) for any treatment group ≤ 5, data for that treatment group will not be displayed at the visit in figure (except the Kaplan-Meier figure), but all data will be included in the corresponding table summary.

# 22. Prior ARV regimen

All subjects will have one of the following prior ARV regimen identified based on ARVs entered in the ARV eCRF: E/C/F/TAF, E/C/F/TDF, ATV+RTV+FTC/TDF.

Use ARV dataset and include all prior and/or current ARVs (ARV.CMSCAT = 'Prior ARV' or 'Current ARV') with taken on or up to 2 days prior to the randomized phase first dose date meeting the following criteria:

| If CMTRT contains Only the specified ARVs: | Re-code as follows for baseline regimen |
|---|---|
| E/C/F/TAF | |
| GENVOYA | E/C/F/TAF |
| NRTI/INI: GENVOYA (EVG+COBI+FTC+TAF) | |
| EVG/COBI/FTC/TDF | E/C/F/TDF |
| NRTI/INI: STRIBILD (EVG+COBI+FTC+TDF) | E/C/F/1DF |
| ATAZANAVIR/RITONAVIR+FTC+TDF | |
| ATV/R+FTC/TDF | |
| NRTI: TRUVADA (FTC+TDF) or PI: ATAZANAVIR (ATV) or PI: RITONAVIR (RTV) | ATV+RTV+FTC/TDF |
| TDF/FTC/ATV/R | |

#### 23. HIV/HBV and HIV/HCV Coinfection:

• The following table presents the HBV and HCV tests with all possible values. Values that have an asterisk after them denote a "positive" (or "quantifiable" for HBV DNA and HCV RNA) result while all others denote a "negative" result.

| Label | LBTESTCD | LBTEST | Possible Values |
|---|---|---|---|
| HBsAg | CNT63 | Hep B Surface Ag | "Positive"*, "Positive, Confirmed"*, "Negative" |
| HBsAg | ATT2 | Hep. B Surf. Ag Qual(-70)-PS | "Repeat reactive, confirmed"*, "Repeat Reactive Unconfirmed", "Non-Reactive" |
| HBsAb | CNT353 | anti-Hep B Surface Ag2<br>Qual | "Positive"*, "Negative" |
| HBcAb | CNT68 | Hepatitis B Core Total | "Positive"*, "Negative" |
| HBV DNA | GET1883 | HBV DNA CAP/CTM<br>2.0-EDTA-CL | "No HBV DNA detected", "<20 IU/mL HBV DNA detected", ">170000000"*, NUMERICAL VALUE when < 29 IU/mL, NUMERICAL VALUE when ≥ 29 IU/nL * |
| HCVAb | CNT350 | Hepatitis C Virus<br>Antibody | "Positive"*, "Indeterminate", "Negative" |
| HCVAb | CNT458 | Hepatitis C<br>AntibodyEDTApl-CL | "Positive"*, "Indeterminate", "Negative" |
| HCV RNA | GET1881 | HCV RNA CAP/CTM<br>2.0EDTA-CL | "No HCV RNA detected", "<15 IU/mL HCV RNA detected", NUMERICAL VALUE* |

- For baseline coinfection, when considering the different laboratory tests, take the latest, non-missing record on or prior to the first dose date for each test (eg, HBsAg, HBsAb, HBcAb, and HBV DNA)
  - o The baseline coinfection status will be one of the three values: Yes/No/Null
  - The following tables provide combinations of HBV and HCV tests and the corresponding baseline coinfection status

| HBsAg | HBsAb | HBcAb | HBV DNA | <b>Coinfection Status</b> |
|---|---|---|---|---|
| Positive | - | - | - | Y |
| Negative | Positive | - | - | N |
| | Negative | Positive | Quantifiable | Y |
| | | | Not Quantifiable | N |
| | | | Missing | Null |
| | | Negative | - | N |
| | | Missing | Quantifiable | Null |
| | | | Not Quantifiable | N |
| | | | Missing | Null |
| | Missing | Positive | Quantifiable | Null |
| | | | Not Quantifiable | N |
| | | | Missing | Null |

| HBsAg | HBsAb | HBcAb | HBV DNA | <b>Coinfection Status</b> |
|---------|----------|----------|------------------|---------------------------|
| | | Negative | - | N |
| | | Missing | Quantifiable | Null |
| | | | Not Quantifiable | N |
| | | | Missing | Null |
| Missing | Positive | - | - | Null |
| | Negative | Positive | Quantifiable | Y |
| | | | Not Quantifiable | Null |
| | | | Missing | Null |
| | | Negative | - | Null |
| | | Missing | - | Null |
| | Missing | - | - | Null |

<sup>&</sup>quot;-" means any value can be present, as it does not affect the classification.

| HCVAb | HCV RNA | Coinfection Status |
|----------|------------------|--------------------|
| Positive | Quantifiable | Y |
| | Not Quantifiable | N |
| | Missing | Null |
| Negative | - | N |
| Missing | Quantifiable | Null |
| | Not Quantifiable | N |
| | Missing | Null |

<sup>&</sup>quot;-" means any value can be present, as it does not affect the classification

- For incident coinfection, all laboratory tests must share the same accession number and if any set of values meets the criteria, then the subject is considered to have incident coinfection
  - o The incident coinfection status will be one of two values: Yes/Null
  - o The following tables provide combinations of HBV and HCV tests that are considered "Y" for incident coinfection status (all others are considered Null)

| HBsAg | HBsAb | HBcAb | HBV DNA | Coinfection Status |
|----------|----------|----------|--------------|--------------------|
| Positive | - | - | - | Y |
| Negative | Negative | Positive | Quantifiable | Y |
| Missing | Negative | Positive | Quantifiable | Y |

| HCVAb | HCV RNA | Coinfection Status |
|-----------|--------------|--------------------|
| Positive* | - | Y |
| - | Quantifiable | Y |

<sup>\*</sup>Subjects with positive HCVAb postbaseline must also have negative or missing HCVAb at baseline in order to be considered as having incident HIV/HCV coinfection.

- For adverse events, the start date must be after the first dose date and on or prior to the last dose date in the randomized phase
- o For incomplete AE start dates, please follow the logic specified in Section 7.1.5.2, but modify the second criterion to read, "The month and year (or year) of the AE onset is the same as or before the month and year (or year) of the date of the last dose of study drug"
- 24. HBV DNA test codes: If the result of the lab test code GET1883 (HBV DNA CAP/CTM 2.0-EDTA-CL) is listed as ">170000000", a reflexive test code GET1884 (HBV DNA CAP/CTM 2.0Dil-EDTA-CL) should be performed and will share the same accession number as the original GET1883 test. In this instance, use the result from GET1884 instead of GET1883 when determining HBV DNA. If reflexive test is not available, HBV DNA level will be determined based on lab test code GET1883.
- 25. Puerto Rico was combined with the United States when we evaluate the treatment effect across countries
- 26. LDL: Conversions between 2<sup>nd</sup> and 3<sup>rd</sup> generations

LDL was analyzed by 2 different assays in the study: 2nd generation (including RCT2394, RCT2312, and RCT2811) and 3rd generation (RCT3870). Samples collected at earlier visits were analyzed using LDL 2nd generation assay. Samples collected at later visits were analyzed using LDL 3rd generation assay. The conversion formulas are as follow:

2nd Gen (mmol/L) = (3rd Gen - 0.0626)/0.882

3rd Gen (mmol/L) =  $(0.882 \times 2nd \text{ Gen}) + 0.0626$ 

For this analysis, since most of the LDL tests were from the 2nd generation, we only requested conversion from 3rd generation to 2nd generation.

For the analysis of change from baseline in fasting direct LDL: the sample analyzed by LDL 3rd generation assay will be converted to 2nd generation as a new record with test codes of LIP.LDL.00.02 in raw data. During ADaM stage, a derived parameter code (FLDL2) for "Fasting LDL Cholesterol 2ND GEN Combined" will be generated to pool the records from both original (including test codes RCT2394, RCT2312, and RCT2811) and converted (LIP.LDL.00.02) 2nd generation results to calculate the change from baseline in fasting direct LDL.

<sup>&</sup>quot;-" means any value can be present, as it does not affect the classification

For the analysis of toxicity grade for fasting direct LDL: toxicity grade will be based on the Gilead grading results (ie, toxgrg) from original values before conversion. In another words, during ADaM stage, a derived parameter code (FLDLTOX) for "Fasting LDL Cholesterol for Toxicity" will be generated to pool the records from 2nd generation (including RCT2394, RCT2312, and RCT2811) and 3rd generation (ie, RCT3870) to derive treatment-emergent toxicity grades, maximum postbaseline toxicity grades, etc.

27. AE action taken for study drug regimen containing multiple pills (eg, ATV + RTV + FTC/TDF) is derived as the most severe actions from all pills in the regimen. The increasing order of severity of AE action taken is: Unknown, Not Applicable, Dose Not Changed, Drug Interrupted, and Drug Withdrawn.